CLINICAL TRIAL: NCT04502693
Title: A Phase III, Randomized, Controlled, Observer-blind Study to Demonstrate Effectiveness, Immunogenicity and Safety of GSK's Meningococcal Group B and Combined ABCWY Vaccines When Administered to Healthy Adolescents and Young Adults
Brief Title: Effectiveness of GlaxoSmithKline Biologicals S.A's Meningococcal Group B and Combined ABCWY Vaccines in Healthy Adolescents and Young Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 205416; 2019-001666-15 (EudraCT Number)
Record Dates: First submitted 2020-08-04; First posted 2020-08-06 (Actual); Results first posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Infections, Meningococcal
Keywords: Bexsero; Menveo; MenABCWY; Effectiveness; Invasive meningococcal disease; Meningitis
MeSH Terms: conditions — Meningococcal Infections; Meningitis | interventions — 4CMenB vaccine; MenACWY; Meningococcal Vaccines; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Observer-blinded study. Recipients & study evaluators will be unaware of vaccine administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (7):
- MenB_0_2_6 Group (Experimental): Participants received 3 doses of rMenB+OMV NZ vaccine on Day 1, Day 61 and Day 181. Participants received 1 dose of MenACWY vaccine at Day 211 as a standard of care.
  Interventions: Combination Product: rMenB+OMV NZ vaccine; Biological: Meningococcal Groups A, C, W and Y Conjugate Vaccine (MenACWY)
- MenB_0_6 Group (Experimental): Participants received 2 doses of rMenB+OMV NZ vaccine on Day 1, and Day 181, 1 dose of MenACWY vaccine on Day 61. Participants received 1 dose of Placebo on Day 211 to maintain blinding.
  Interventions: Combination Product: rMenB+OMV NZ vaccine; Biological: Meningococcal Groups A, C, W and Y Conjugate Vaccine (MenACWY); Combination Product: Placebo
- ABCWY-1 Group (Experimental): Participants received 2 doses of MenABCWY lot 1 vaccine at Day 1 and Day 181 and 2 doses of placebo at Day 61 and Day 211.
  Interventions: Combination Product: Placebo; Combination Product: MenABCWY-1
- ABCWY-2 Group (Experimental): Participants received 2 doses of MenABCWY lot 2 vaccine at Day 1 and Day 181 and 2 doses of placebo at Day 61 and Day 211.
  Interventions: Combination Product: Placebo; Combination Product: MenABCWY-2
- ABCWY-3 Group (Experimental): Participants received 2 doses of MenABCWY lot 3 vaccine at Day 1 and Day 181 and 2 doses of placebo at Day 61 and Day 211.
  Interventions: Combination Product: Placebo; Combination Product: MenABCWY-3
- ACWY Group (Active Comparator): Participants received 1 dose of MenACWY vaccine at Day 1,1 dose of placebo at Day 61 and 1 dose of rMenB+OMV NZ vaccine on Day 181. Participants received 1 dose of rMenB+OMV NZ vaccine on Day 211 as standard of care.
  Interventions: Combination Product: rMenB+OMV NZ vaccine; Biological: Meningococcal Groups A, C, W and Y Conjugate Vaccine (MenACWY); Combination Product: Placebo
- ABCWY_Pooled (Experimental): Participants received 2 doses of either MenABCWY Lot 1, Lot 2, or Lot 3 vaccine on Day 1 and Day 181 and 1 dose of placebo on Day 61. Participants received 1 dose of placebo on Day 211 to maintain blinding.
  To evaluate the effectiveness of 2 doses of the MenABCWY vaccines against rMenB+OMV and MenACWY vaccines, participants from the ABCWY-1, ABCWY-2, and ABCWY-3 groups were pooled into a single group.
  Interventions: Combination Product: MenABCWY-1; Combination Product: MenABCWY-2; Combination Product: MenABCWY-3

INTERVENTIONS:
Combination Product: rMenB+OMV NZ vaccine — rMenB+OMV NZ vaccine was administered intramuscularly.
  Other Names: Bexsero
  Arms: ACWY Group; MenB_0_2_6 Group; MenB_0_6 Group
Biological: Meningococcal Groups A, C, W and Y Conjugate Vaccine (MenACWY) — MenACWY vaccine was administered intramuscularly.
  Other Names: Menveo
  Arms: ACWY Group; MenB_0_2_6 Group; MenB_0_6 Group
Combination Product: Placebo — Placebo was administered intramuscularly.
  Other Names: NaCl, saline solution
  Arms: ABCWY-1 Group; ABCWY-2 Group; ABCWY-3 Group; ACWY Group; MenB_0_6 Group
Combination Product: MenABCWY-1 — Lot 1 of the MenABCWY vaccine was administered intramuscularly.
  Arms: ABCWY-1 Group; ABCWY_Pooled
Combination Product: MenABCWY-2 — Lot 2 of the MenABCWY vaccine was administered intramuscularly.
  Arms: ABCWY-2 Group; ABCWY_Pooled
Combination Product: MenABCWY-3 — Lot 3 of the MenABCWY vaccine was administered intramuscularly.
  Arms: ABCWY-3 Group; ABCWY_Pooled

SUMMARY:
The purpose of this study was to evaluate the effectiveness of 2 doses or 3 doses of GSK's licenced meningococcal group B Bexsero (rMenB+OMV NZ) vaccine and of 2 doses of GSK's investigational combined meningococcal (MenABCWY) vaccine (GSK3536819A) in healthy adolescents and young adults. The immunogenicity and safety were evaluated in the study.

DETAILED DESCRIPTION:
As per the feedback from the Center for Biologics Evaluation and Research (CBER), the scope of this post-marketing commitment study was extended to demonstrate the effectiveness, immunogenicity, and safety of GSK's investigational combined meningococcal ABCWY vaccine along with the rMenB+OMV NZ vaccine. Note that the rMenB+OMV and MenACWY vaccines provided to the MenB_0_2_6, MenB_0_6 group, and MenACWY group, respectively, at day 211 were only as part of the standard care of treatment and to maintain blinding. These vaccination schedules were not considered for any endpoint evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Subjects or/and subjects' parent(s)/Legally Acceptable Representative(s) [LAR(s)] who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written or witnessed/thumb printed informed consent obtained from the subject/parent(s)/LAR(s) of the subject prior to performance of any study specific procedure.
* Written informed assent obtained from the subject (if applicable) prior to performing any study specific procedure.
* A male or female between, and including, 10 and 25 years of age (i.e. 25 years + 364 days) at the time of the first vaccination.
* Healthy subjects as established by medical history physical examination and clinical judgment of the investigator before entering into the study.
* Subjects who are either unvaccinated with MenACWY vaccine or have received a single previous dose of MenACWY vaccine can participate in the study, if they have received it at least 4 years prior to informed consent and assent as applicable (with the exception of meningococcal C vaccination, if the last dose of MenC was received at ≤24 months of age).
* Female subjects of non-childbearing potential may be enrolled in the study. Non-childbearing potential is defined as pre-menarche, current bilateral tubal ligation or occlusion, hysterectomy, bilateral ovariectomy or post-menopause*.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception until 30 days after completion of Visit 6.

    * A female is considered to be of non-childbearing potential prior to menarche and after natural or induced menopause. Natural menopause is recognized to have occurred after 12 consecutive months of amenorrhea for which there is no other obvious pathological or physiological cause. Induced menopause is recognized to have occurred after hysterectomy, after bilateral oophorectomy, or iatrogenic ablation of ovarian function.

Exclusion Criteria:

Medical conditions

* Current or previous, confirmed or suspected disease caused by N. meningitidis.
* Household contact with and/or intimate exposure to an individual with laboratory confirmed N. meningitidis infection within 60 days of enrolment.
* Progressive, unstable or uncontrolled clinical conditions.
* Clinical conditions representing a contraindication to intramuscular vaccination and blood draws.
* Any neuroinflammatory, congenital neurological conditions, encephalopathies, seizures. History of febrile convulsions should not lead to exclusion.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine(s)/product(s).

  * Hypersensitivity, including allergy, to any component of vaccines, including diphtheria toxoid (CRM 197) and latex medicinal products or medical equipment whose use is foreseen in this study.
* Abnormal function or modification of the immune system resulting from:

  * Autoimmune disorders or immunodeficiency syndromes.
  * Systemic administration of corticosteroids (PO/IV/IM) for more than 14 consecutive days within 90 days prior to study vaccination until the post-vaccination 3 blood sample (Visit 6). This will mean prednisone - ≥20 mg/day (for adult subjects) or ≥0.5 mg/kg/day (for paediatric subjects), or equivalent. Inhaled and topical steroids are allowed.
  * Administration of antineoplastic and immunomodulating agents or radiotherapy within 90 days prior to study vaccination.
  * Administration of long-acting immune-modifying drugs at any time during the study period (e.g. infliximab).
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.

Prior/Concomitant therapy

* Use of any investigational or non-registered product other than the study vaccine(s)/product(s) during the period starting 30 days before the first dose of study vaccine(s)/product(s) (Day -29 to Day 1), or planned use during the study period.
* Previous vaccination against any group B meningococcal vaccine at any time prior to informed consent and assent as applicable.
* Administration of immunoglobulins and/or any blood products or plasma derivatives during the period starting 90 days before the first dose of study vaccine/ product or planned administration during the study period until the post-vaccination 3 blood sample (Visit 6).
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs during the period starting 90 days prior to the vaccine/product dose(s) until the post-vaccination 3 blood sample (Visit 6). For corticosteroids, this will mean prednisone ≥20 mg/day (for adult subjects) or ≥0.5 mg/kg/day (for paediatric subjects), or equivalent. Inhaled and topical steroids are allowed.

Prior/Concurrent clinical study experience

• Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product.

Other exclusions

* Child in care.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* History of /current chronic alcohol abuse and/or drug abuse as determined by the investigator.
* Any study personnel or immediate dependants, family, or household member.

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3657 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (98):
- United States (54):
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Glendale, Arizona
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Bell Gardens, California
  - GSK Investigational Site, Canoga Park, California
  - GSK Investigational Site, Garden Grove, California
  - GSK Investigational Site, Inglewood, California
  - GSK Investigational Site, Los Gatos, California
  - GSK Investigational Site, Cutler Bay, Florida
  - GSK Investigational Site, Lake City, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Oviedo, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Adairsville, Georgia
  - GSK Investigational Site, Buford, Georgia
  - GSK Investigational Site, Columbus, Georgia
  - GSK Investigational Site, Hinesville, Georgia
  - GSK Investigational Site, Nampa, Idaho
  - GSK Investigational Site, Oak Brook, Illinois
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Bardstown, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Beverly, Massachusetts
  - GSK Investigational Site, Fall River, Massachusetts
  - GSK Investigational Site, Grosse Pointe Woods, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Petal, Mississippi
  - GSK Investigational Site, Missoula, Montana
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Grants Pass, Oregon
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, North Charleston, South Carolina
  - GSK Investigational Site, West Columbia, South Carolina
  - GSK Investigational Site, Laredo, Texas
  - GSK Investigational Site, Plano, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Kaysville, Utah
  - GSK Investigational Site, Layton, Utah
  - GSK Investigational Site, Murray, Utah
  - GSK Investigational Site, Orem, Utah
  - GSK Investigational Site, Roy, Utah
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, South Jordan, Utah
  - GSK Investigational Site, Syracuse, Utah
  - GSK Investigational Site, Falls Church, Virginia
  - GSK Investigational Site, Newport News, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Suffolk, Virginia
  - GSK Investigational Site, Cheney, Washington
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Marshfield, Wisconsin
- Australia (7):
  - GSK Investigational Site, Sydney, New South Wales
  - GSK Investigational Site, Gold Coast, Queensland
  - GSK Investigational Site, Taringa, Queensland
  - GSK Investigational Site, Tarragindi, Queensland
  - GSK Investigational Site, Geelong, Victoria
  - GSK Investigational Site, Melbourne, Victoria
  - GSK Investigational Site, Nedlands, Western Australia
- Canada (11):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Sarnia, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Pointe-Claire, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Québec
- Czechia (11):
  - GSK Investigational Site, České Budejovice
  - GSK Investigational Site, České Budějovice
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Jindřichův Hradec
  - GSK Investigational Site, Kladno
  - GSK Investigational Site, Mělník
  - GSK Investigational Site, Pardubice
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Příbram
  - GSK Investigational Site, Trutnov
  - GSK Investigational Site, Týnec nad Sázavou
- GSK Investigational Site, Tallinn, Estonia
- Finland (9):
  - GSK Investigational Site, Espoo
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Jarvenpaa
  - GSK Investigational Site, Kokkola
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Pori
  - GSK Investigational Site, Seinäjoki
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
- Turkey (Türkiye) (5):
  - GSK Investigational Site, Adana
  - GSK Investigational Site, Ankara
  - GSK Investigational Site, Eskişehir
  - GSK Investigational Site, Izmir
  - GSK Investigational Site, Kayseri

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.

REFERENCES:
- [Derived] Nolan T, Bhusal C, Beran J, Bloch M, Cetin BS, Dinleyici EC, Drazan D, Kokko S, Koski S, Laajalahti O, Langley JM, Ramet M, Richmond PC, Silas P, Tapiero B, Tiong F, Tipton M, Ukkonen B, Ulukol B, Lattanzi M, Trapani M, Willemsen A, Toneatto D; QUINTET study group. Breadth of immune response, immunogenicity, reactogenicity, and safety for a pentavalent meningococcal ABCWY vaccine in healthy adolescents and young adults: results from a phase 3, randomised, controlled observer-blinded trial. Lancet Infect Dis. 2025 May;25(5):560-573. doi: 10.1016/S1473-3099(24)00667-4. Epub 2024 Dec 5. PMID 39647494

RESULTS

PARTICIPANT FLOW:
Recruitment Details: As pre-specified in protocol:
  * Participant flow, Baseline characteristics, Effectiveness and immunogenicity data are presented for MenB_0_2_6 group, MenB_0_6 group, ACWY group, ABCWY pooled group.
  * Lot-to-lot consistency analysis data are presented for individual ABCWY lot groups (ABCWY-1, ABCWY-2 and ABCWY-3) as Lot-to-Lot assessment was limited to the objective on lot-to-lot consistency only.
Pre-assignment Details: Out of 3657 participants enrolled,19 participants did not receive vaccination as they did not meet the eligibility criteria, therefore only 3638 participants were included in the Exposed Set and started the study.
Period: Overall Study
Arm/Group | MenB_0_2_6 Group | MenB_0_6 Group | ABCWY_Pooled | ACWY Group
Started | 897 | 906 | 1657 | 178
ABCWY-1 Group | 0 | 0 | 549 | 0
ABCWY-2 Group | 0 | 0 | 554 | 0
ABCWY-3 Group | 0 | 0 | 554 | 0
Completed | 797 | 811 | 1497 | 163
Not Completed | 100 | 95 | 160 | 15
Not completed — Adverse Event | 7 | 6 | 11 | 1
Not completed — Lost to Follow-up | 32 | 36 | 69 | 4
Not completed — Protocol Violation | 8 | 8 | 16 | 1
Not completed — Withdrawal by Subject | 46 | 38 | 54 | 7
Not completed — MIGRATED / MOVED FROM THE STUDY AREA | 6 | 7 | 9 | 1
Not completed — Other | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: As pre-specified in the protocol, data reported in the Baseline characteristics are presented for MenB_0_2_6 group, MenB_0_6 group, ACWY group, ABCWY pooled group.
Groups:
- Total: Total of all reporting groups
Arm/Group | MenB_0_2_6 Group | MenB_0_6 Group | ABCWY_Pooled | ACWY Group | Total
Number analyzed (Participants) | 897 | 906 | 1657 | 178 | 3638
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.5 (4.7) | 16.5 (4.7) | 16.5 (4.7) | 16.9 (4.6) | 16.5 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 464 | 446 | 933 | 100 | 1943
  Male | 433 | 460 | 724 | 78 | 1695
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 5 | 3 | 0 | 13
  Asian | 43 | 60 | 71 | 9 | 183
  Black or African American | 33 | 29 | 59 | 6 | 127
  Native Hawaiian or Other Pacific Islander | 3 | 1 | 3 | 0 | 7
  White | 796 | 791 | 1492 | 162 | 3241
  Other, Unspecified | 17 | 20 | 29 | 1 | 67

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Blood Samples Without Bactericidal Serum Activity Against Each of the Endemic US N. Meningitidis Serogroup B Strains at 1 Month After the 3-dose (0,2,6-M), 2-dose(0,6-M) Vaccination Schedule of rMenB+OMV and 1 Dose of MenACWY
Description: The effectiveness (test-based) of rMenB+OMV vaccine at 1 month after the 3 doses in MenB_0_2_6 group and 1 month after the 2 dose schedule in MenB_0_6 group when compared to one dose of MenACWY vaccination in ACWY group, against a panel of N. meningitidis serogroup B strains was measured in terms of percentage of samples without bactericidal activity using endogenous complement human Serum Bactericidal Assay (enc-hSBA), which provides a qualitative assessment (yes/no) of the presence of sufficient bactericidal antibodies in human sera to kill a meningococcal strain at a specific dilution of 1:4.
  Participants were randomly selected for testing against each strain therefore only a subset of participants were tested for each of the strains.
Time Frame: At 1 month after vaccination schedule (i.e., Day 211 for MenB_0_2_6 group [3-dose schedule] and MenB_0_6 group, and Day 31 for ACWY group)
Population: Analysis was performed on blood samples collected from Per Protocol Set (PPS) ,which included participants who received at least 1 dose of the study treatment to which they were randomized and have post-vaccination data for the specified analysis at the specified timepoints and did not have any protocol deviations that lead to exclusion from the PPS.
  Number of Participants analyzed = Total number of participants included in PPS.
Measure: Number; unit: Percentage of blood samples
Units Other Than Participants: Samples
Arm/Group | MenB_0_2_6 Group | MenB_0_6 Group | ACWY Group
Number analyzed (Participants) | 740 | 751 | 147
Number analyzed (Samples) | 25596 | 26142 | 4374
Percentage of blood samples | 13.3 | 14.4 | 79
Statistical Analysis 1: Comparison: MenB_0_2_6 Group vs ACWY Group; To demonstrate the effectiveness of the rMenB+OMV NZ vaccine against a randomly selected panel of endemic US N. meningitidis serogroup B invasive disease strains as measured by bactericidal activity using enc-hSBA at 1 month after the 3-dose (0,2,6-months) schedule in MenB_0_2_6 group when compared to 1 month after the MenACWY dose in the ACWY group; Test type: Other — Effectiveness of rMenB+OMV NZ vaccine is demonstrated if the LL of the 2-sided 97.5% CI for Vaccine Effectiveness (VE) against the selected strain panel between the MenB_0_2_6 and the ACWY groups is above 65%. VE is defined as 1- Risk Ratio (RR) = (1- percentage of samples without bactericidal serum activity at 1:4 dilution in MenB group / percentage of samples without bactericidal serum activity at 1:4 dilution in the ACWY group) x100 percentage; VE (Vaccine Effectiveness) = 83.2, 97.5% CI 2-sided [81.9 to 84.4]
Statistical Analysis 2: Comparison: MenB_0_6 Group vs ACWY Group; To demonstrate the effectiveness of the rMenB+OMV NZ vaccine against a randomly selected panel of endemic US N. meningitidis serogroup B invasive disease strains as measured by bactericidal activity using enc-hSBA at 1 month after the 2-dose (0,6-M) schedule in MenB_0_6 group when compared to 1 month after the MenACWY dose in the ACWY group; Test type: Other — Effectiveness of rMenB+OMV NZ vaccine is demonstrated if the LL of the 2-sided 97.5% CI for VE against the selected strain panel between the MenB_0_ 6 and the ACWY groups is above 65%. VE is defined as 1- RR = (1- percentage of samples without bactericidal serum activity at 1:4 dilution in MenB group / percentage of samples without bactericidal serum activity at 1:4 dilution in the ACWY group) x100 percentage; VE = 81.8, 97.5% CI 2-sided [80.4 to 83.1]

2. Primary Outcome: Percentage of Blood Samples Without Bactericidal Serum Activity Against Each of the Endemic US N. Meningitidis Serogroup B Strains at 1 Month After the 2-dose (0,2-M) Vaccination Schedule of rMenB+OMV and 1 Dose of MenACWY
Description: The effectiveness (test-based) of rMenB+OMV vaccine at 1 month after the 2 doses in MenB_0_2_6 group when compared to one dose of MenACWY vaccination in ACWY group, against a panel of N. meningitidis serogroup B strains was measured in terms of percentage of samples without bactericidal activity using endogenous complement human Serum Bactericidal Assay (enc-hSBA), which provides a qualitative assessment (yes/no) of the presence of sufficient bactericidal antibodies in human sera to kill a meningococcal strain at a specific dilution of 1:4.
  Participants were randomly selected for testing against each strain therefore only a subset of participants were tested for each of the strains.
Time Frame: At 1 month after vaccination schedule (i.e., Day 91 for the MenB_0_2_6 group [2-dose schedule] and Day 31 for ACWY group)
Population: Analysis was performed on blood samples collected from Per Protocol Set (PPS) ,which included participants who received at least 1 dose of the study treatment to which they were randomized and have post-vaccination data for the specific analysis at specified timepoints and did not have any protocol deviations that lead to exclusion from the PPS.
  Number of Participants analyzed = Total number of participants included in PPS.
Measure: Number; unit: Percentage of blood samples
Units Other Than Participants: Samples
Arm/Group | MenB_0_2_6 Group | ACWY Group
Number analyzed (Participants) | 740 | 147
Number analyzed (Samples) | 27569 | 4374
Percentage of blood samples | 16.8 | 79
Statistical Analysis 1: Comparison: MenB_0_2_6 Group vs ACWY Group; To demonstrate the effectiveness of the rMenB+OMV NZ vaccine against a randomly selected panel of endemic US N. meningitidis serogroup B invasive disease strains as measured by bactericidal activity using enc-hSBA at 1 month after the 2-dose (0,2-M) schedule in MenB_0_2_6 group when compared to 1 month after the MenACWY dose in the ACWY group; Test type: Other — Effectiveness of rMenB+OMV NZ vaccine is demonstrated if the LL of the 2-sided 97.5% CI for VE against the selected strain panel between the MenB_0_2_6 and the ACWY groups is above 65%. VE is defined as 1- RR = (1- percentage of samples without bactericidal serum activity at 1:4 dilution in MenB group / percentage of samples without bactericidal serum activity at 1:4 dilution in the ACWY group) x100 percentage; VE = 78.7, 97.5% CI 2-sided [77.2 to 80.1]

3. Primary Outcome: Percentage of Participants Whose Sera Kill Greater Than or Equal to (>=) 70% of the Strains Tested Using Enc-hSBA at 1 Month After the 3-dose (0,2,6-M) Schedule of rMenB+OMV and 2-dose(0,6-M) Schedule of rMenB+OMV
Description: The effectiveness (responder-based) of the rMenB+OMV NZ vaccine was measured in terms of percentage of participants whose sera kill >=70% of the strains tested using enc-hSBA, calculated based on Clopper Pearson method. Effectiveness is demonstrated if Lower Limit (LL) of the two-sided 97.5% CI for the percentages of participants whose sera kill ≥70% of strains is above 65%.
Time Frame: At 1 month after vaccination schedule (i.e., Day 211 for MenB_0_2_6 group [3-dose schedule] and MenB_0_6 group)
Population: Analysis was performed on the Full Analysis Set, which included participants who were randomized, received at least 1 dose of the study treatment and had post-vaccination effectiveness available for the specified analysis at the specified timepoint.
Measure: Number (97.5% Confidence Interval); unit: Percentage of participants
Arm/Group | MenB_0_2_6 Group | MenB_0_6 Group
Number analyzed (Participants) | 790 | 813
Percentage of participants | 93.4 (91.2) [91.2 to 95.2] | 89.8 (87.2) [87.2 to 92]

4. Primary Outcome: Percentage of Participants Whose Sera Kill >=70% of the Strains Tested Using Enc-hSBA at 1 Month After the 2-dose (0,2-M) Schedule of rMenB+OMV
Description: as for outcome 3
Time Frame: At 1 month after vaccination schedule (i.e., Day 91 for the MenB_0_2_6 group [2-dose schedule])
Population: as for outcome 3
Measure: Number (97.5% Confidence Interval); unit: Percentage of participants
Arm/Group | MenB_0_2_6 Group
Number analyzed (Participants) | 831
Percentage of participants | 84.8 (81.8) [81.8 to 87.5]

5. Primary Outcome: Geometric Mean Titers (GMTs) Against Serogroups A, C, W and Y for Each Lot (ABCWY-1 Group, ABCWY-2 Group and ABCWY-3 Group) at 1 Month After the Last Vaccination of MenABCWY
Description: Immune response was measured in terms of hSBA GMTs directed against serogroups A, C, W and Y. As pre-specified in the protocol, the data reported in this outcome measures data were presented for individual lots to demonstrate the consistency of the immune response of 3 lots (ABCWY- 1 Group, ABCWY-2 Group, and ABCWY-3 Group) of the ACWY component of the MenABCWY vaccine.
Time Frame: At 1 month after the last vaccination of MenABCWY (Day 211)
Population: Analysis was performed on Per Protocol Set (PPS), which included participants who received at least 1 dose of the study treatment to which they were randomized and have post-vaccination data for the specified analysis at specified timepoints and did not have any protocol deviations that lead to exclusion from the PPS.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | ABCWY-1 Group | ABCWY-2 Group | ABCWY-3 Group
Number analyzed (Participants) | 452 | 449 | 458
Titers
  Men A: number analyzed (Participants) | 448 | 443 | 454
  Men A | 336.4 [299.3 to 378.0] | 349.9 [311.5 to 393.0] | 390.4 [347.4 to 438.8]
  Men C: number analyzed (Participants) | 448 | 449 | 456
  Men C | 1036.7 [877.6 to 1224.5] | 1130.2 [958.1 to 1333.4] | 888.4 [752.1 to 1049.2]
  Men W | 564.5 [497.9 to 639.9] | 635.5 [561.0 to 719.9] | 640.1 [564.6 to 725.6]
  Men Y: number analyzed (Participants) | 451 | 449 | 457
  Men Y | 536.7 [464.5 to 620.2] | 623.9 [540.4 to 720.2] | 644.3 [557.6 to 744.6]
Statistical Analysis 1: Comparison: ABCWY-1 Group vs ABCWY-2 Group; To demonstrate lot-to-lot consistency of the immune responses of ABCWY-1 and ABCWY-2 lots of the MenACWY component of the MenABCWY vaccine, as measured by hSBA GMTs directed against serogroup A at 1 month after last vaccination (Day 211); Test type: Equivalence — Lot-to-lot consistency is claimed if the 2-sided 95% CIs for the ratio of hSBA GMTs of antibodies against each of the serogroups A, C, W and Y are within the [0.5;2.0] equivalence interval for each pair of lots; GMT ratio = 0.96, 95% CI 2-sided [0.84 to 1.10]
Statistical Analysis 2: Comparison: ABCWY-1 Group vs ABCWY-3 Group; To demonstrate lot-to-lot consistency of the immune responses of ABCWY-1 and ABCWY-3 lots of the MenACWY component of the MenABCWY vaccine, as measured by hSBA GMTs directed against serogroup A at 1 month after last vaccination (Day 211); Test type: Equivalence — Lot-to-lot consistency is claimed if the 2-sided 95% CIs for the ratio of hSBA GMTs of antibodies against each of the serogroups A, C, W and Y is within the [0.5;2.0] equivalence interval for each pair of lots; GMT ratio = 0.86, 95% CI 2-sided [0.75 to 0.98]
Statistical Analysis 3: Comparison: ABCWY-2 Group vs ABCWY-3 Group; To demonstrate lot-to-lot consistency of the immune responses of ABCWY-2 and ABCWY-3 lots of the MenACWY component of the MenABCWY vaccine, as measured by hSBA GMTs directed against serogroup A at 1 month after last vaccination (Day 211); Test type: Equivalence — [test comment as in outcome 5, analysis 2]; GMT ratio = 0.90, 95% CI 2-sided [0.78 to 1.02]
Statistical Analysis 4: Comparison: ABCWY-1 Group vs ABCWY-2 Group; To demonstrate lot-to-lot consistency of the immune responses of ABCWY-1 and ABCWY-2 lots of the MenACWY component of the MenABCWY vaccine, as measured by hSBA GMTs directed against serogroup C at 1 month after last vaccination (Day 211); Test type: Equivalence — [test comment as in outcome 5, analysis 1]; GMT ratio = 0.92, 95% CI 2-sided [0.76 to 1.11]
Statistical Analysis 5: Comparison: ABCWY-1 Group vs ABCWY-3 Group; To demonstrate lot-to-lot consistency of the immune responses of ABCWY-1 and ABCWY-3 lots of the MenACWY component of the MenABCWY vaccine, as measured by hSBA GMTs directed against serogroup C at 1 month after last vaccination (Day 211); Test type: Equivalence — [test comment as in outcome 5, analysis 2]; GMT ratio = 1.17, 95% CI 2-sided [0.97 to 1.41]
Statistical Analysis 6: Comparison: ABCWY-2 Group vs ABCWY-3 Group; To demonstrate lot-to-lot consistency of the immune responses of ABCWY-2 and ABCWY-3 lots of the MenACWY component of the MenABCWY vaccine, as measured by hSBA GMTs directed against serogroup C at 1 month after last vaccination (Day 211); Test type: Equivalence — [test comment as in outcome 5, analysis 2]; GMT ratio = 1.27, 95% CI 2-sided [1.05 to 1.54]
Statistical Analysis 7: Comparison: ABCWY-1 Group vs ABCWY-2 Group; To demonstrate lot-to-lot consistency of the immune responses of ABCWY-1 and ABCWY-2 lots of the MenACWY component of the MenABCWY vaccine, as measured by hSBA GMTs directed against serogroup W at 1 month after last vaccination (Day 211); Test type: Equivalence — [test comment as in outcome 5, analysis 1]; GMT ratio = 0.89, 95% CI 2-sided [0.77 to 1.02]
Statistical Analysis 8: Comparison: ABCWY-1 Group vs ABCWY-3 Group; To demonstrate lot-to-lot consistency of the immune responses of ABCWY-1 and ABCWY-3 lots of the MenACWY component of the MenABCWY vaccine, as measured by hSBA GMTs directed against serogroup W at 1 month after last vaccination (Day 211); Test type: Equivalence — [test comment as in outcome 5, analysis 2]; GMT ratio = 0.88, 95% CI 2-sided [0.77 to 1.02]
Statistical Analysis 9: Comparison: ABCWY-2 Group vs ABCWY-3 Group; To demonstrate lot-to-lot consistency of the immune responses of ABCWY-2 and ABCWY-3 lots of the MenACWY component of the MenABCWY vaccine, as measured by hSBA GMTs directed against serogroup W at 1 month after last vaccination (Day 211); Test type: Equivalence — [test comment as in outcome 5, analysis 2]; GMT ratio = 0.99, 95% CI 2-sided [0.86 to 1.14]
Statistical Analysis 10: Comparison: ABCWY-1 Group vs ABCWY-2 Group; To demonstrate lot-to-lot consistency of the immune responses of ABCWY-1 and ABCWY-2 lots of the MenACWY component of the MenABCWY vaccine, as measured by hSBA GMTs directed against serogroup Y at 1 month after last vaccination (Day 211); Test type: Equivalence — [test comment as in outcome 5, analysis 1]; GMT ratio = 0.86, 95% CI 2-sided [0.73 to 1.01]
Statistical Analysis 11: Comparison: ABCWY-1 Group vs ABCWY-3 Group; To demonstrate lot-to-lot consistency of the immune responses of ABCWY-1 and ABCWY-3 lots of the MenACWY component of the MenABCWY vaccine, as measured by hSBA GMTs directed against serogroup Y at 1 month after last vaccination (Day 211); Test type: Equivalence — [test comment as in outcome 5, analysis 2]; GMT ratio = 0.83, 95% CI 2-sided [0.71 to 0.98]
Statistical Analysis 12: Comparison: ABCWY-2 Group vs ABCWY-3 Group; To demonstrate lot-to-lot consistency of the immune responses of ABCWY-2 and ABCWY-3 lots of the MenACWY component of the MenABCWY vaccine, as measured by hSBA GMTs directed against serogroup Y at 1 month after last vaccination (Day 211); Test type: Equivalence — [test comment as in outcome 5, analysis 2]; GMT ratio = 0.97, 95% CI 2-sided [0.82 to 1.14]

6. Primary Outcome: Percentage of Participants With 4-fold Rise in hSBA Titers Against N. Meningitidis Serogroups A, C, W and Y at 1 Month After Last MenABCWY Vaccination (Pooled Lots) and MenACWY Vaccination (for the ACWY Group), Relative to Baseline
Description: Four-fold rise is defined as: If the pre-vaccination hSBA titer is < 4, then post-vaccination hSBA titer should be >= 16 . If the pre-vaccination hSBA titer is >= limit of detection (LOD) but < LL of quantification (LLOQ), then post-vaccination hSBA titer should be >= 4 times the LLOQ. If the pre-vaccination hSBA titer is >= LLOQ, then post-vaccination hSBA titer should be >= 4 times the pre-vaccination hSBA titer.
  As pre-specified in the protocol, data reported in this outcome measure were presented for ACWY group, ABCWY pooled group to evaluate the immunological non-inferiority of 2 doses of the MenABCWY vaccines against MenACWY vaccines, participants from the ABCWY-1, ABCWY-2, and ABCWY-3 groups were pooled into a single group.
Time Frame: At 1 month after vaccination schedule (i.e., Day 211 for the ABCWY_Pooled group and Day 31 for the ACWY Group) compared to Day 1 (baseline)
Population: Analysis was performed on Per Protocol Set, which included participants who received at least 1 dose of the study treatment to which they were randomized and have post-vaccination data for the specified analysis at specified timepoints and did not have any protocol deviations that lead to exclusion from the PPS.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ABCWY_Pooled | ACWY Group
Number analyzed (Participants) | 1196 | 119
Percentage of participants
  Men A: number analyzed (Participants) | 1170 | 112
  Men A | 97.0 [95.9 to 97.9] | 85.7 [77.8 to 91.6]
  Men C: number analyzed (Participants) | 1189 | 114
  Men C | 97.2 [96.1 to 98.1] | 50.0 [40.5 to 59.5]
  Men W: number analyzed (Participants) | 1185 | 115
  Men W | 97.0 [95.9 to 97.9] | 61.7 [52.2 to 70.6]
  Men Y | 96.7 [95.6 to 97.7] | 69.7 [60.7 to 77.8]
Statistical Analysis 1: Comparison: ABCWY_Pooled vs ACWY Group; To demonstrate the immunological non-inferiority of the MenABCWY vaccine compared to the MenACWY vaccine in participants without a previous MenACWY vaccination (unprimed) as measured by the percentages of participants, achieving a 4-fold rise in hSBA titers against N. meningitidis serogroup A at 1 month after the last MenABCWY vaccination (Day 211) and 1 month after the MenACWY vaccination; Test type: Non-Inferiority — Non-inferiority of MenABCWY vaccine is demonstrated if the LL of the 2-sided 95% CI for the difference in percentage of participants with 4-fold rise between the 2 groups is above -10%; Difference in percentage of participants; Difference in percentage of participants = 11.29, 95% CI 2-sided [5.88 to 19.01]
Statistical Analysis 2: Comparison: ABCWY_Pooled vs ACWY Group; To demonstrate the immunological non-inferiority of the MenABCWY vaccine compared to the MenACWY vaccine in participants without a previous MenACWY vaccination (unprimed) as measured by the percentages of participants, achieving a 4-fold rise in hSBA titers against N. meningitidis serogroup C at 1 month after the last MenABCWY vaccination (Day 211) and 1 month after the MenACWY vaccination; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; Difference in percentage of participants = 47.22, 95% CI 2-sided [38.14 to 56.30]
Statistical Analysis 3: Comparison: ABCWY_Pooled vs ACWY Group; To demonstrate the immunological non-inferiority of the MenABCWY vaccine compared to the MenACWY vaccine in participants without a previous MenACWY vaccination (unprimed) as measured by the percentages of participants, achieving a 4-fold rise in hSBA titers against N. meningitidis serogroup W at 1 month after the last MenABCWY vaccination (Day 211) and 1 month after the MenACWY vaccination; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; Difference in percentage of participants = 35.31, 95% CI 2-sided [26.88 to 44.49]
Statistical Analysis 4: Comparison: ABCWY_Pooled vs ACWY Group; To demonstrate the immunological non-inferiority of the MenABCWY vaccine compared to the MenACWY vaccine in participants without a previous MenACWY vaccination (unprimed) as measured by the percentages of participants, achieving a 4-fold rise in hSBA titers against N. meningitidis serogroup Y at 1 month after the last MenABCWY vaccination (Day 211) and 1 month after the MenACWY vaccination; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; Difference in percentage of participants = 26.99, 95% CI 2-sided [19.38 to 35.81]

7. Primary Outcome: Percentage of Blood Samples Without Bactericidal Serum Activity Against Each of the Endemic U.S N. Meningitidis Serogroup B Strains at 1 Month After Last MenABCWY Vaccination (Pooled Lots) and MenACWY Vaccination (for the ACWY Group)
Description: The effectiveness (test-based) of 2 doses of MenABCWY vaccine when compared to 1 dose of MenACWY vaccine, against a panel of N. meningitidis serogroup B strains was measured in terms of percentage of samples without bactericidal activity using enc-hSBA, which provides a qualitative assessment (yes/no) of the presence of sufficient bactericidal antibodies in human sera to kill a meningococcal strain at a specific dilution of 1:4.
  As pre-specified in the protocol, data reported in this outcome measure were presented for ACWY group and ABCWY pooled group to evaluate the effectiveness of 2 doses of the MenABCWY vaccines against MenACWY vaccines, participants from the ABCWY-1, ABCWY-2, and ABCWY-3 groups were pooled into a single group.
Time Frame: At 1 month after the vaccination schedule (i.e., Day 211 for the ABCWY_Pooled group and Day 31 for the ACWY group)
Population: Analysis was performed on blood samples collected from Per Protocol Set (PPS), which included participants who received at least 1 dose of the study treatment to which they were randomized and have post-vaccination data for the specified analysis at specified timepoints and did not have any protocol deviations that lead to exclusion from the PPS.
Measure: Number; unit: Percentage of blood samples
Units Other Than Participants: Samples
Arm/Group | ABCWY_Pooled | ACWY Group
Number analyzed (Participants) | 1356 | 147
Number analyzed (Samples) | 25715 | 4374
Percentage of blood samples | 17.4 | 79
Statistical Analysis 1: Comparison: ABCWY_Pooled vs ACWY Group; To demonstrate the effectiveness of the MenABCWY vaccine against a randomly selected panel of endemic US N. meningitidis serogroup B invasive disease strains as measured by enc-hSBA at 1 month after the last MenABCWY vaccination (Day 211) when compared to 1 month after the MenACWY vaccination; Test type: Other — Effectiveness of MenABCWY vaccine is demonstrated if the LL of the 2-sided 95% CI for VE against the selected strain panel between the ABCWY and the ACWY groups is above 65%. VE is defined as 1- RR = (1- percentage of samples without bactericidal serum activity at 1:4 dilution in ABCWY_Pooled group / percentage of samples without bactericidal serum activity at 1:4 dilution in the ACWY group) x100 percentage; VE = 77.9, 95% CI 2-sided [76.6 to 79.2]

8. Primary Outcome: Percentage of Blood Samples With Bactericidal Serum Activity Against Each of the Endemic U.S N. Meningitidis Serogroup B Strains at 1 Month After the Last MenABCWY Dose (Pooled Lots) and 2-dose(0,2-M) Schedule of rMenB+OMV
Description: The effectiveness was measured in terms of percentage of samples with bactericidal activity using enc-hSBA, which provides a qualitative assessment (yes/no) of the presence of sufficient bactericidal antibodies in human sera to kill a meningococcal strain at a specific dilution of 1:4. As pre-specified in the protocol, data reported in this outcome measure were presented for MenB_0_2_6 Group and ABCWY pooled group to evaluate the effectiveness of 2 doses of the MenABCWY vaccines against MenACWY vaccines, participants from the ABCWY-1, ABCWY-2, and ABCWY-3 groups were pooled into a single group.
Time Frame: At 1 month after the vaccination schedule (i.e., Day 211 for the ABCWY_Pooled group and Day 91 for the MenB_0_2_6 Group [2-dose schedule])
Population: Analysis was performed on blood samples collected from PPS, which included participants who received at least 1 dose of the study treatment to which they were randomized and have post-vaccination data for the specified analysis at specified timepoints and did not have any protocol deviations that lead to exclusion from the PPS.
Measure: Number; unit: Percentage of blood samples
Units Other Than Participants: Samples
Arm/Group | MenB_0_2_6 Group | ABCWY_Pooled
Number analyzed (Participants) | 740 | 1356
Number analyzed (Samples) | 27569 | 25715
Percentage of blood samples | 83.1 | 82.5
Statistical Analysis 1: Comparison: MenB_0_2_6 Group vs ABCWY_Pooled; To demonstrate the non-inferiority of the effectiveness of the MenABCWY vaccine (0,6-months schedule) compared to the rMenB+OMV NZ vaccine (0,2-months) in terms of percentage of samples with bactericidal serum activity using enc-hSBA against a randomly selected panel of endemic US N. meningitidis serogroup B invasive disease strains; Test type: Non-Inferiority — Non-inferiority of MenABCWY to rMenB+OMV NZ is demonstrated if LL of the 2-sided 95% CI for the difference in percentages of samples with bactericidal serum activity at 1:4 dilution is above -5%; Difference in percentage of participants = -0.61, 95% CI 2-sided [-1.25 to 0.03]

9. Primary Outcome: Percentage of Participants Whose Sera Kill >=70% of the Strains Tested Using Enc-hSBA at 1 Month After the Last Vaccination in the ABCWY Group (Pooled Lots)
Description: The effectiveness (responder-based) of the MenABCWY vaccine is measured in terms of percentage of participants whose sera kill >=70% of the strains tested using enc-hSBA, being calculated based on Clopper Pearson method. Effectiveness is demonstrated Lower Limit (LL) of the two-sided 97.5% CI for the percentages of participants whose sera kill ≥70% of strains tested for MenABCWY is above 65%.
Time Frame: At 1 month after the last vaccination of MenABCWY (Day 211)
Population: Analysis was performed on the FAS, which included all participants who were randomized, received at least 1 dose of the study treatment, and had post-vaccination effectiveness data available for the specified analysis at the specified time points.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ABCWY_Pooled
Number analyzed (Participants) | 817
Percentage of participants | 84.1 (81.4) [81.4 to 86.5]

10. Primary Outcome: Number of Participants With Any Solicited Local Adverse Events (AEs) After the First Study Intervention Administration
Description: Assessed solicited local adverse events were injection or administration site = pain, erythema, swelling, induration. Any = occurrence of the adverse event regardless of intensity grade. Any erythema and swelling = adverse event reported with a surface diameter greater than 0 millimeters. No solicited AEs were collected after vaccination on Day 211 because these vaccines were administered as part of standard of care and to maintain blinding. As pre- specified in the protocol, data reported in this outcome measure were presented for MenB_0_2_6 group, MenB_0_6 group, ACWY group, ABCWY pooled group.
Time Frame: During 7 days after the first study intervention administration occurring at Day 1
Population: Analysis was performed on the Solicited Safety Set (SSS), which included participants who received at least 1 dose of the study treatment and had solicited safety data during the specified period.
Measure: Count of Participants; unit: Participants
Arm/Group | MenB_0_2_6 Group | MenB_0_6 Group | ABCWY_Pooled | ACWY Group
Number analyzed (Participants) | 885 | 894 | 1638 | 178
Participants
  Pain | 807 | 819 | 1503 | 67
  Erythema | 90 | 86 | 216 | 11
  Swelling | 87 | 89 | 217 | 11
  Induration | 60 | 64 | 150 | 7

11. Primary Outcome: Number of Participants With Any Solicited Local Adverse Events (AEs) After the Second Study Intervention Administration
Description: Assessed solicited local adverse events were injection or administration site pain, erythema, swelling, induration. Any = occurrence of the adverse event regardless of intensity grade. Any erythema and swelling = adverse event reported with a surface diameter greater than 0 millimeters. No solicited AEs were collected after vaccination on Day 211 because these vaccines were administered as part of standard of care and to maintain blinding. As pre- specified in the protocol, data reported in this outcome measure were presented for MenB_0_2_6 group, MenB_0_6 group, ACWY group, ABCWY pooled group.
Time Frame: During 7 days after the second study intervention administration occurring at Day 61
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | MenB_0_2_6 Group | MenB_0_6 Group | ABCWY_Pooled | ACWY Group
Number analyzed (Participants) | 823 | 813 | 1511 | 161
Participants
  Pain | 714 | 224 | 205 | 30
  Erythema | 89 | 26 | 5 | 1
  Swelling | 99 | 22 | 5 | 1
  Induration | 67 | 19 | 6 | 0

12. Primary Outcome: Number of Participants With Any Solicited Local Adverse Events (AEs) After the Third Study Intervention Administration
Description: as for outcome 11
Time Frame: During 7 days after the third study intervention administration occurring at Day 181
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | MenB_0_2_6 Group | MenB_0_6 Group | ABCWY_Pooled | ACWY Group
Number analyzed (Participants) | 765 | 759 | 1428 | 148
Participants
  Pain | 677 | 676 | 1258 | 126
  Erythema | 118 | 87 | 168 | 11
  Swelling | 107 | 85 | 176 | 13
  Induration | 52 | 57 | 114 | 12

13. Primary Outcome: Number of Participants With Any Solicited Systemic AEs After the First Study Intervention Administration
Description: Assessed solicited systemic AEs were fatigue, nausea, myalgia, arthralgia, headache and fever [temperature >= 38.0°C]. Any = occurrence of the adverse event regardless of intensity grade or relation to study vaccination. No solicited AEs were collected after vaccination on Day 211 because these vaccines were administered as part of standard of care and to maintain blinding. As pre- specified in the protocol, data reported in this outcome measure were presented for MenB_0_2_6 group, MenB_0_6 group, ACWY group, ABCWY pooled group.
Time Frame: During 7 days after the first study intervention administration occurring at Day 1
Population: Analysis was performed on the Solicited Safety Set (SSS), which included participants who receive at least 1 dose of the study treatment and had solicited safety data during the specified period.
Measure: Count of Participants; unit: Participants
Arm/Group | MenB_0_2_6 Group | MenB_0_6 Group | ABCWY_Pooled | ACWY Group
Number analyzed (Participants) | 885 | 894 | 1638 | 178
Participants
  Fatigue | 423 | 414 | 828 | 78
  Nausea | 112 | 111 | 242 | 27
  Myalgia | 92 | 106 | 242 | 13
  Arthralgia | 56 | 70 | 133 | 17
  Headache | 358 | 330 | 681 | 69
  Fever (C) | 19 | 17 | 55 | 3

14. Primary Outcome: Number of Participants With Any Solicited Systemic AEs After the Second Study Intervention Administration
Description: as for outcome 13
Time Frame: During 7 days after the second study intervention administration occurring at Day 61
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | MenB_0_2_6 Group | MenB_0_6 Group | ABCWY_Pooled | ACWY Group
Number analyzed (Participants) | 823 | 813 | 1511 | 161
Participants
  Fatigue | 372 | 228 | 345 | 36
  Nausea | 104 | 56 | 85 | 18
  Myalgia | 110 | 46 | 55 | 3
  Arthralgia | 72 | 332.0 | 35 | 6
  Headache | 301 | 223 | 332 | 31
  Fever (C) | 22 | 12 | 18 | 1

15. Primary Outcome: Number of Participants With Any Solicited Systemic AEs After the Third Study Intervention Administration
Description: as for outcome 13
Time Frame: During 7 days after the third study intervention administration occurring at Day 181
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | MenB_0_2_6 Group | MenB_0_6 Group | ABCWY_Pooled | ACWY Group
Number analyzed (Participants) | 765 | 759 | 1428 | 148
Participants
  Fatigue | 374 | 341 | 602 | 56
  Nausea | 94 | 84 | 147 | 14
  Myalgia | 106 | 109 | 168 | 17
  Arthralgia | 71 | 53 | 104 | 7
  Headache | 302 | 284 | 509 | 39
  Fever (C) | 21 | 23 | 27 | 2

16. Primary Outcome: Number of Participants With Any Unsolicited AEs After the First Study Intervention Administration
Description: Unsolicited AEs are defined as any AE reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms were reported as an unsolicited AE. Any Unsolicited AEs (including Serious adverse events (SAEs), AEs leading to withdrawal, Adverse event of special interest (AESIs) and medically attended AEs were collected during 30 days after vaccination 1-3. For vaccination on Day 211 (Vaccination 4), conducted as part of standard of care and to maintain blinding, no eDiary data or all unsolicited AEs were collected for the 30 days following vaccination. However, SAEs, AEs leading to withdrawal, AESIs and medically attended AEs were collected throughout study duration. As pre-specified in the protocol, data reported in this outcome measure were presented for MenB_0_2_6 group, MenB_0_6 group, ACWY group, ABCWY pooled group.
Time Frame: During the 30 days after the first study intervention administration occurring at Day 1
Population: Analysis was performed on the Unsolicited Safety Set (USS), which included participants who received at least 1 dose of the study treatment and had Unsolicited safety data during the specified period.
Measure: Count of Participants; unit: Participants
Arm/Group | MenB_0_2_6 Group | MenB_0_6 Group | ABCWY_Pooled | ACWY Group
Number analyzed (Participants) | 893 | 900 | 1648 | 178
Participants | 90 | 124 | 217 | 29

17. Primary Outcome: Number of Participants With Any Unsolicited AEs After the Second Study Intervention Administration
Description: as for outcome 16
Time Frame: During the 30 days after the second study intervention administration occurring at Day 61
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | MenB_0_2_6 Group | MenB_0_6 Group | ABCWY_Pooled | ACWY Group
Number analyzed (Participants) | 851 | 855 | 1579 | 170
Participants | 106 | 88 | 160 | 15

18. Primary Outcome: Number of Participants With Any Unsolicited AEs After the Third Study Intervention Administration
Description: as for outcome 16
Time Frame: During the 30 days after the third study intervention administration occurring at Day 181
Population: Analysis was performed on the Unsolicited Safety Set (USS), which included all participants who received at least 1 dose of the study treatment and had Unsolicited safety data during the specified period.
Measure: Count of Participants; unit: Participants
Arm/Group | MenB_0_2_6 Group | MenB_0_6 Group | ABCWY_Pooled | ACWY Group
Number analyzed (Participants) | 815 | 823 | 1521 | 166
Participants | 96 | 94 | 183 | 19

19. Primary Outcome: Number of Participants With SAEs, AEs Leading to Withdrawal, AESIs and Medically Attended AEs
Description: A SAEs is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity and is a congenital anomaly/birth defect in the offspring of a study subject. AESIs are predefined (serious or non-serious) AEs of scientific and medical concern specific to the product or program, for which ongoing monitoring and rapid communication by the investigator to the sponsor can be appropriate, because such an event might warrant further investigation to characterize and understand it. Medically attended AEs are symptoms or illnesses requiring hospitalization, or emergency room visit, or visit to/by a health care provider. As pre-specified in the protocol, data reported in this outcome measure were presented for MenB_0_2_6 group, MenB_0_6 group, ACWY group, ABCWY pooled group.
Time Frame: Throughout the study period (Day 1 to Day 361)
Population: Analysis was performed on the Unsolicited Safety Set (USS), which included participants who received at least 1 dose of the study treatment and report unsolicited AEs/report not having unsolicited AEs.
Measure: Count of Participants; unit: Participants
Arm/Group | MenB_0_2_6 Group | MenB_0_6 Group | ABCWY_Pooled | ACWY Group
Number analyzed (Participants) | 893 | 900 | 1648 | 178
Participants
  SAEs | 20 | 22 | 25 | 5
  AEs leading to withdrawal | 6 | 4 | 4 | 1
  AESIs | 1 | 1 | 6 | 0
  medically attended AEs | 238 | 288 | 479 | 44

20. Secondary Outcome: Percentage of Participants With 4-fold Rise in hSBA Titers Against N.Meningitidis Group B Strains at 1 Month After Last MenABCWY Dose(ABCWY Group-pooled Lots) and 1 Month After 2-dose(0,2-M) Schedule of rMenB+OMV NZ Relative to Baseline
Description: The immunogenicity is measured as percentage of participants achieving a 4-fold rise in hSBA titers against N. meningitidis serogroup B indicator strains (M14459, 96217, M13520 and NZ98/254 for fHbp, NadA, NHBA and PorA P1.4 antigens, respectively). 4-fold rise per each indicator strain was defined as a post-vaccination hSBA titre ≥16 for participants with a pre-vaccination hSBA titre <4; a post-vaccination hSBA titre ≥4 times the LLOQ for participants with a pre-vaccination hSBA titre ≥LOD and <LLOQ; a post-vaccination hSBA titre ≥4 times the pre-vaccination hSBA titre for participants with a pre-vaccination hSBA titre ≥ LLOQ. As pre-specified in the protocol, data reported in this outcome measure were presented for MenB_0_2_6 Group and ABCWY pooled group to evaluate the effectiveness of 2 doses of the MenABCWY vaccines against MenACWY vaccines, participants from the ABCWY-1, ABCWY-2, and ABCWY-3 groups were pooled into a single group.
Time Frame: At 1 month after the vaccination schedule (i.e., Day 211 for the ABCWY_Pooled group and Day 91 for the MenB_0_2_6 Group [2-dose schedule]) compared to Day 1 (Baseline)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MenB_0_2_6 Group | ABCWY_Pooled
Number analyzed (Participants) | 719 | 678
Percentage of participants
  fHbp (M14459) Ab: number analyzed (Participants) | 719 | 675
  fHbp (M14459) Ab | 74.7 [71.3 to 77.8] | 79.7 [76.5 to 82.7]
  NadA (96217) Ab: number analyzed (Participants) | 717 | 671
  NadA (96217) Ab | 96.4 [94.7 to 97.6] | 92.7 [90.5 to 94.5]
  NHBA (M13520) Ab: number analyzed (Participants) | 718 | 678
  NHBA (M13520) Ab | 58.6 [54.9 to 62.3] | 61.9 [58.2 to 65.6]
  PorA (NZ98/254) Ab: number analyzed (Participants) | 704 | 642
  PorA (NZ98/254) Ab | 53.3 [49.5 to 57.0] | 42.2 [38.4 to 46.1]

21. Secondary Outcome: Percentage of Blood Samples Without Bactericidal Serum Activity Against Each of the Endemic U.S N. Meningitidis Serogroup B Strains at 1 Month After the Last MenABCWY Dose and 3-dose (0,2,6-M), 2-dose(0,6-M) Schedule of rMenB+OMV and 1 Dose of MenACWY
Description: The effectiveness of the 3 dose (0,2,6-M) and 2 dose (0,6-M ) schedule of rMenB+OMV NZ vaccine and 2 doses of MenABCWY vaccine when compared to 1 month after the MenACWY vaccination (Day 31), against a panel of N. meningitidis serogroup B strains is measured in terms of percentage of samples without bactericidal activity using enc-hSBA, which provides a qualitative assessment (yes/no) of the presence of sufficient bactericidal antibodies in human sera to kill a meningococcal strain at a specific dilution of 1:4. As pre-specified in the protocol, data reported in this outcome measure were presented for the MenB_0_2_6 group, MenB_0_6 group,ACWY group and ABCWY pooled group, participants from the ABCWY-1, ABCWY-2, and ABCWY-3 groups were pooled into a single group.
Time Frame: At 1 month after the vaccination schedule (i.e., Day 211 for the MenB_0_2_6 group [3 dose schedule], MenB_0_6 group, ABCWY_Pooled group and Day 31 for the MenACWY group)
Population: Analysis was performed on blood samples collected from FAS, which included participants who were randomized, received at least one dose of the study treatment, and had post-vaccination effectiveness data available for the specified analysis at the specified time points. Participants were randomly selected for testing against each strain therefore only a subset of participants were tested for each of the strains.
  Number of Participants analyzed = Total number of participants included in FAS.
Measure: Number; unit: Percentage of blood samples
Units Other Than Participants: Samples
Arm/Group | MenB_0_2_6 Group | MenB_0_6 Group | ABCWY_Pooled | ACWY Group
Number analyzed (Participants) | 790 | 813 | 817 | 136
Number analyzed (Samples) | 281 | 282 | 288 | 58
Percentage of blood samples
  Meningitis B M10713 Ab: number analyzed (Samples) | 252 | 247 | 251 | 45
  Meningitis B M10713 Ab | 0.4 | 0.4 | 1.2 | 15.6
  Meningitis B M08641 Ab: number analyzed (Samples) | 229 | 259 | 237 | 29
  Meningitis B M08641 Ab | 6.6 | 6.2 | 8.0 | 96.6
  Meningitis B M12898 Ab: number analyzed (Samples) | 242 | 265 | 249 | 41
  Meningitis B M12898 Ab | 8.4 | 11.4 | 12.1 | 68.1
  Meningitis B M09150 Ab: number analyzed (Samples) | 249 | 222 | 273 | 36
  Meningitis B M09150 Ab | 5.2 | 8.5 | 12.6 | 73.0
  Meningitis B M09401 Ab: number analyzed (Samples) | 243 | 275 | 288 | 49
  Meningitis B M09401 Ab | 50.2 | 46.5 | 57 | 98.0
  Meningitis B M07463 Ab: number analyzed (Samples) | 259 | 274 | 256 | 49
  Meningitis B M07463 Ab | 1.5 | 1.8 | 3.5 | 49
  Meningitis B M10496 Ab: number analyzed (Samples) | 263 | 261 | 257 | 47
  Meningitis B M10496 Ab | 54.4 | 47.9 | 68.9 | 100.0
  Meningitis B M14530 Ab: number analyzed (Samples) | 241 | 257 | 284 | 37
  Meningitis B M14530 Ab | 2.1 | 1.6 | 3.2 | 100.0
  Meningitis B M15668 Ab: number analyzed (Samples) | 237 | 270 | 262 | 49
  Meningitis B M15668 Ab | 0.8 | 2.2 | 0.8 | 87.8
  Meningitis B M14028 Ab: number analyzed (Samples) | 246 | 282 | 283 | 37
  Meningitis B M14028 Ab | 2.8 | 5.7 | 4.9 | 100
  Meningitis B M09909 Ab: number analyzed (Samples) | 244 | 265 | 261 | 42
  Meningitis B M09909 Ab | 79.1 | 83.4 | 86.2 | 100.0
  Meningitis B M14385 Ab: number analyzed (Samples) | 235 | 237 | 259 | 43
  Meningitis B M14385 Ab | 0.9 | 0.8 | 0.0 | 16.3
  Meningitis B M07992 Ab: number analyzed (Samples) | 237 | 252 | 274 | 36
  Meningitis B M07992 Ab | 0.4 | 0.0 | 0.4 | 0.0
  Meningitis B M09155 Ab: number analyzed (Samples) | 234 | 255 | 230 | 45
  Meningitis B M09155 Ab | 1.7 | 2.0 | 1.3 | 97.8
  Meningitis B M13085 Ab: number analyzed (Samples) | 256 | 253 | 255 | 44
  Meningitis B M13085 Ab | 13.5 | 27.5 | 26.6 | 69.3
  Meningitis B M18303 Ab: number analyzed (Samples) | 241 | 252 | 264 | 40
  Meningitis B M18303 Ab | 2.9 | 4.0 | 9.5 | 100.0
  Meningitis B M18711 Ab: number analyzed (Samples) | 252 | 237 | 262 | 33
  Meningitis B M18711 Ab | 5.2 | 4.2 | 9.5 | 75.8
  Meningitis B M15009 Ab: number analyzed (Samples) | 262 | 254 | 242 | 37
  Meningitis B M15009 Ab | 11.8 | 20.5 | 31.8 | 86.5
  Meningitis B M07773 Ab: number analyzed (Samples) | 269 | 262 | 251 | 35
  Meningitis B M07773 Ab | 0.7 | 0.4 | 0.4 | 74.3
  Meningitis B M09662 Ab: number analyzed (Samples) | 267 | 266 | 255 | 48
  Meningitis B M09662 Ab | 61.4 | 50.8 | 66.3 | 95.8
  Meningitis B M18483 Ab: number analyzed (Samples) | 228 | 233 | 222 | 37
  Meningitis B M18483 Ab | 3.0 | 5.1 | 3.7 | 72.2
  Meningitis B M11906 Ab: number analyzed (Samples) | 264 | 271 | 260 | 39
  Meningitis B M11906 Ab | 23.7 | 30.3 | 39.9 | 84.7
  Meningitis B M14987 Ab: number analyzed (Samples) | 250 | 274 | 270 | 35
  Meningitis B M14987 Ab | 1.2 | 8.8 | 12.7 | 68.6
  Meningitis B M12014 Ab: number analyzed (Samples) | 249 | 270 | 254 | 46
  Meningitis B M12014 Ab | 0.4 | 0.7 | 1.2 | 67.4
  Meningitis B M18200 Ab: number analyzed (Samples) | 228 | 247 | 242 | 47
  Meningitis B M18200 Ab | 6.3 | 14.8 | 14.9 | 33.7
  Meningitis B M08912 Ab: number analyzed (Samples) | 225 | 247 | 237 | 40
  Meningitis B M08912 Ab | 0.4 | 0.0 | 0.0 | 0.0
  Meningitis B M16748 Ab: number analyzed (Samples) | 262 | 252 | 260 | 45
  Meningitis B M16748 Ab | 0.8 | 0.0 | 0 | 0.0
  Meningitis B M08152 Ab: number analyzed (Samples) | 208 | 215 | 223 | 35
  Meningitis B M08152 Ab | 22.4 | 25.3 | 32.8 | 66.8
  Meningitis B M09973 Ab: number analyzed (Samples) | 252 | 270 | 247 | 48
  Meningitis B M09973 Ab | 0.8 | 1.1 | 3.0 | 83.3
  Meningitis B M15352 Ab: number analyzed (Samples) | 237 | 249 | 245 | 33
  Meningitis B M15352 Ab | 8.9 | 8.4 | 17.8 | 97.0
  Meningitis B M15165 Ab: number analyzed (Samples) | 249 | 250 | 240 | 42
  Meningitis B M15165 Ab | 0.0 | 1.2 | 2.1 | 92.9
  Meningitis B M08127 Ab: number analyzed (Samples) | 269 | 250 | 287 | 51
  Meningitis B M08127 Ab | 0.7 | 0.4 | 0.7 | 84.3
  Meningitis B M18347 Ab: number analyzed (Samples) | 234 | 262 | 239 | 44
  Meningitis B M18347 Ab | 45.4 | 50.9 | 51.8 | 82.1
  Meningitis B M12500 Ab: number analyzed (Samples) | 223 | 253 | 241 | 43
  Meningitis B M12500 Ab | 0.9 | 2.4 | 2.5 | 95.3
  Meningitis B M07499 Ab: number analyzed (Samples) | 242 | 251 | 256 | 51
  Meningitis B M07499 Ab | 70.7 | 75.7 | 80.1 | 100.0
  Meningitis B M09960 Ab: number analyzed (Samples) | 243 | 247 | 251 | 33
  Meningitis B M09960 Ab | 1.2 | 0 | 0 | 3.0
  Meningitis B M18045 Ab: number analyzed (Samples) | 236 | 251 | 272 | 41
  Meningitis B M18045 Ab | 0 | 0.4 | 0 | 92.7
  Meningitis B M10548 Ab: number analyzed (Samples) | 234 | 243 | 261 | 58
  Meningitis B M10548 Ab | 8.1 | 11.9 | 12.5 | 74.1
  Meningitis B M09354 Ab: number analyzed (Samples) | 246 | 240 | 241 | 40
  Meningitis B M09354 Ab | 1.2 | 1.3 | 0 | 80.0
  Meningitis B M11051 Ab: number analyzed (Samples) | 246 | 282 | 247 | 46
  Meningitis B M11051 Ab | 61.0 | 64.2 | 66.7 | 97.8
  Meningitis B M10104 Ab: number analyzed (Samples) | 247 | 241 | 239 | 41
  Meningitis B M10104 Ab | 58.7 | 52.3 | 63.5 | 97.6
  Meningitis B M13361 Ab: number analyzed (Samples) | 258 | 268 | 250 | 34
  Meningitis B M13361 Ab | 0.8 | 0.4 | 0.4 | 85.3
  Meningitis B M11042 Ab: number analyzed (Samples) | 217 | 249 | 254 | 43
  Meningitis B M11042 Ab | 19.8 | 25.5 | 33.5 | 85.7
  Meningitis B M18467 Ab: number analyzed (Samples) | 255 | 223 | 250 | 47
  Meningitis B M18467 Ab | 1.2 | 0.4 | 0.8 | 78.7
  Meningitis B M11113 Ab: number analyzed (Samples) | 255 | 253 | 269 | 51
  Meningitis B M11113 Ab | 30.1 | 39.5 | 49.5 | 75.2
  Meningitis B M07253 Ab: number analyzed (Samples) | 260 | 245 | 255 | 40
  Meningitis B M07253 Ab | 34.7 | 33.8 | 50.2 | 86.4
  Meningitis B M07356 Ab: number analyzed (Samples) | 235 | 235 | 266 | 29
  Meningitis B M07356 Ab | 0.4 | 0 | 1.1 | 41.4
  Meningitis B M10710 Ab: number analyzed (Samples) | 254 | 253 | 270 | 40
  Meningitis B M10710 Ab | 1.6 | 2.0 | 1.4 | 92.5
  Meningitis B M17147 Ab: number analyzed (Samples) | 261 | 279 | 214 | 41
  Meningitis B M17147 Ab | 2.3 | 5.4 | 2.3 | 100
  Meningitis B M14401 Ab: number analyzed (Samples) | 241 | 266 | 253 | 43
  Meningitis B M14401 Ab | 1.7 | 0.4 | 1.2 | 83.7
  Meningitis B M14293 Ab: number analyzed (Samples) | 251 | 247 | 224 | 47
  Meningitis B M14293 Ab | 45.8 | 25.1 | 45.2 | 95.7
  Meningitis B M08540 Ab: number analyzed (Samples) | 258 | 261 | 222 | 34
  Meningitis B M08540 Ab | 1.6 | 0.8 | 0 | 38.2
  Meningitis B M07960 Ab: number analyzed (Samples) | 277 | 241 | 241 | 39
  Meningitis B M07960 Ab | 3.6 | 4.1 | 1.8 | 94.9
  Meningitis B M16135 Ab: number analyzed (Samples) | 254 | 230 | 257 | 41
  Meningitis B M16135 Ab | 0 | 1.7 | 0.8 | 95.1
  Meningitis B M14548 Ab: number analyzed (Samples) | 267 | 266 | 274 | 38
  Meningitis B M14548 Ab | 2.6 | 3.4 | 3.2 | 94.7
  Meningitis B M09181 Ab: number analyzed (Samples) | 228 | 276 | 240 | 43
  Meningitis B M09181 Ab | 0 | 0.4 | 0.4 | 72.1
  Meningitis B M14224 Ab: number analyzed (Samples) | 248 | 279 | 277 | 40
  Meningitis B M14224 Ab | 0.4 | 0.4 | 0 | 82.5
  Meningitis B M07452 Ab: number analyzed (Samples) | 260 | 260 | 245 | 47
  Meningitis B M07452 Ab | 2.7 | 8.1 | 17.1 | 85.1
  Meningitis B M13520 Ab: number analyzed (Samples) | 217 | 222 | 242 | 30
  Meningitis B M13520 Ab | 3.2 | 0.9 | 0 | 66.7
  Meningitis B M09385 Ab: number analyzed (Samples) | 228 | 252 | 265 | 32
  Meningitis B M09385 Ab | 0.4 | 1.6 | 0 | 46.9
  Meningitis B M14881 Ab: number analyzed (Samples) | 240 | 278 | 277 | 40
  Meningitis B M14881 Ab | 4.2 | 5.8 | 10 | 95
  Meningitis B M13252 Ab: number analyzed (Samples) | 279 | 241 | 262 | 50
  Meningitis B M13252 Ab | 0.7 | 1.2 | 0.4 | 98
  Meningitis B M07818 Ab: number analyzed (Samples) | 232 | 244 | 228 | 43
  Meningitis B M07818 Ab | 0.4 | 0.8 | 1.3 | 90.7
  Meningitis B M09914 Ab: number analyzed (Samples) | 281 | 257 | 258 | 49
  Meningitis B M09914 Ab | 85.4 | 86.8 | 88.3 | 98
  Meningitis B M15083 Ab: number analyzed (Samples) | 231 | 262 | 241 | 40
  Meningitis B M15083 Ab | 51.4 | 56.7 | 61 | 84.5
  Meningitis B M11290 Ab: number analyzed (Samples) | 264 | 266 | 221 | 34
  Meningitis B M11290 Ab | 61.4 | 61.7 | 67.4 | 100
  Meningitis B M14988 Ab: number analyzed (Samples) | 241 | 269 | 246 | 40
  Meningitis B M14988 Ab | 0.4 | 0 | 1.2 | 60
  Meningitis B M10536 Ab: number analyzed (Samples) | 228 | 223 | 260 | 36
  Meningitis B M10536 Ab | 19.7 | 14.3 | 14.3 | 91.7
  Meningitis B M08959 Ab: number analyzed (Samples) | 252 | 241 | 258 | 47
  Meningitis B M08959 Ab | 0.8 | 0.4 | 1.9 | 85.1
  Meningitis B M08785 Ab: number analyzed (Samples) | 251 | 249 | 260 | 39
  Meningitis B M08785 Ab | 0.8 | 0.4 | 0.4 | 53.8
  Meningitis B M07245 Ab: number analyzed (Samples) | 238 | 248 | 230 | 43
  Meningitis B M07245 Ab | 0 | 0 | 0.9 | 23.3
  Meningitis B M19315 Ab: number analyzed (Samples) | 262 | 254 | 255 | 34
  Meningitis B M19315 Ab | 3.8 | 3.1 | 9.5 | 79.4
  Meningitis B M14376 Ab: number analyzed (Samples) | 234 | 220 | 222 | 41
  Meningitis B M14376 Ab | 0 | 1.4 | 0 | 92.7
  Meningitis B M08994 Ab: number analyzed (Samples) | 226 | 253 | 233 | 31
  Meningitis B M08994 Ab | 2.5 | 7.6 | 6.9 | 62.7
  Meningitis B M11646 Ab: number analyzed (Samples) | 241 | 224 | 250 | 36
  Meningitis B M11646 Ab | 0 | 1.3 | 2 | 83.3
  Meningitis B M13362 Ab: number analyzed (Samples) | 259 | 228 | 231 | 49
  Meningitis B M13362 Ab | 0 | 0.4 | 0.4 | 81.6
  Meningitis B M08080 Ab: number analyzed (Samples) | 236 | 247 | 242 | 45
  Meningitis B M08080 Ab | 27.4 | 41 | 51.6 | 85.7
  Meningitis B M08370 Ab: number analyzed (Samples) | 265 | 262 | 251 | 43
  Meningitis B M08370 Ab | 2.3 | 1.5 | 3.7 | 97.7
  Meningitis B M08129 Ab: number analyzed (Samples) | 245 | 254 | 257 | 28
  Meningitis B M08129 Ab | 4.1 | 4.7 | 7 | 71.4
  Meningitis B M07111 Ab: number analyzed (Samples) | 231 | 254 | 270 | 33
  Meningitis B M07111 Ab | 0.4 | 1.2 | 0.7 | 90.9
  Meningitis B M07537 Ab: number analyzed (Samples) | 241 | 242 | 263 | 47
  Meningitis B M07537 Ab | 95.9 | 95.9 | 97.7 | 100
  Meningitis B M13438 Ab: number analyzed (Samples) | 255 | 262 | 282 | 50
  Meningitis B M13438 Ab | 1.2 | 0.8 | 0 | 16
  Meningitis B M10661 Ab: number analyzed (Samples) | 246 | 275 | 273 | 33
  Meningitis B M10661 Ab | 2 | 2.9 | 2.9 | 97
  Meningitis B M10920 Ab: number analyzed (Samples) | 247 | 252 | 275 | 34
  Meningitis B M10920 Ab | 29.1 | 27.8 | 37.8 | 91.2
  Meningitis B M15564 Ab: number analyzed (Samples) | 240 | 273 | 263 | 40
  Meningitis B M15564 Ab | 0.4 | 0.7 | 0.8 | 77.5
  Meningitis B M10934 Ab: number analyzed (Samples) | 273 | 241 | 256 | 36
  Meningitis B M10934 Ab | 0.4 | 0.8 | 0.8 | 100
  Meningitis B M09400 Ab: number analyzed (Samples) | 254 | 281 | 279 | 39
  Meningitis B M09400 Ab | 0.8 | 1.8 | 0.4 | 97.4
  Meningitis B M08781 Ab: number analyzed (Samples) | 221 | 258 | 229 | 28
  Meningitis B M08781 Ab | 71.9 | 74.4 | 78.2 | 100
  Meningitis B M09173 Ab: number analyzed (Samples) | 238 | 249 | 247 | 42
  Meningitis B M09173 Ab | 0.4 | 0.4 | 0.8 | 95.2
  Meningitis B M14113 Ab: number analyzed (Samples) | 228 | 255 | 264 | 42
  Meningitis B M14113 Ab | 15.4 | 21.2 | 22 | 100
  Meningitis B M08389 Ab: number analyzed (Samples) | 254 | 259 | 250 | 45
  Meningitis B M08389 Ab | 10.7 | 7 | 11.7 | 87.2
  Meningitis B M16822 Ab: number analyzed (Samples) | 239 | 233 | 264 | 34
  Meningitis B M16822 Ab | 67.8 | 76.4 | 82.2 | 100
  Meningitis B M10995 Ab: number analyzed (Samples) | 268 | 258 | 239 | 47
  Meningitis B M10995 Ab | 5.2 | 17.8 | 30.6 | 85.1
  Meningitis B M08780 Ab: number analyzed (Samples) | 236 | 259 | 260 | 40
  Meningitis B M08780 Ab | 1.3 | 0.8 | 1.5 | 92.5
  Meningitis B M09910 Ab: number analyzed (Samples) | 247 | 246 | 257 | 43
  Meningitis B M09910 Ab | 1.6 | 1.2 | 1.2 | 93
  Meningitis B M08320 Ab: number analyzed (Samples) | 262 | 238 | 253 | 45
  Meningitis B M08320 Ab | 33.6 | 39.7 | 43.3 | 87
  Meningitis B M14879 Ab: number analyzed (Samples) | 239 | 242 | 247 | 47
  Meningitis B M14879 Ab | 2.1 | 2.1 | 6.1 | 21.3
  Meningitis B M09345 Ab: number analyzed (Samples) | 251 | 257 | 282 | 48
  Meningitis B M09345 Ab | 19.3 | 20.1 | 33.4 | 81.2
  Meningitis B M14594 Ab: number analyzed (Samples) | 245 | 241 | 238 | 44
  Meningitis B M14594 Ab | 20.8 | 27.4 | 41.2 | 97.7
  Meningitis B M07621 Ab: number analyzed (Samples) | 251 | 260 | 263 | 40
  Meningitis B M07621 Ab | 1.2 | 1.2 | 1.1 | 77.5
  Meningitis B M13568 Ab: number analyzed (Samples) | 261 | 264 | 253 | 40
  Meningitis B M13568 Ab | 5.4 | 3.8 | 3.9 | 95
  Meningitis B M18017 Ab: number analyzed (Samples) | 246 | 247 | 258 | 31
  Meningitis B M18017 Ab | 0.4 | 0 | 1.6 | 96.8
  Meningitis B M08420 Ab: number analyzed (Samples) | 243 | 255 | 256 | 40
  Meningitis B M08420 Ab | 0.8 | 0.4 | 1.6 | 95
  Meningitis B M07959 Ab: number analyzed (Samples) | 236 | 237 | 254 | 35
  Meningitis B M07959 Ab | 1.7 | 2.5 | 1.7 | 97.1
  Meningitis B M06970 Ab: number analyzed (Samples) | 236 | 261 | 253 | 32
  Meningitis B M06970 Ab | 19.6 | 17.6 | 30.2 | 85.7
  Meningitis B M10491 Ab: number analyzed (Samples) | 239 | 262 | 227 | 39
  Meningitis B M10491 Ab | 5.4 | 8.4 | 17 | 82.1
  Meningitis B M13569 Ab: number analyzed (Samples) | 221 | 243 | 247 | 31
  Meningitis B M13569 Ab | 0.9 | 2.9 | 1.2 | 96.8
  Meningitis B M10182 Ab: number analyzed (Samples) | 229 | 234 | 256 | 44
  Meningitis B M10182 Ab | 0.4 | 0 | 0 | 0
  Meningitis B M13547 Ab: number analyzed (Samples) | 251 | 258 | 238 | 44
  Meningitis B M13547 Ab | 2.4 | 7 | 4.7 | 47.7
  Meningitis B M15276 Ab: number analyzed (Samples) | 231 | 231 | 259 | 41
  Meningitis B M15276 Ab | 0.4 | 0 | 1.5 | 87.8

22. Secondary Outcome: Percentage of Blood Samples Without Bactericidal Serum Activity Using Enc-hSBA Against Each of the Endemic U.S N. Meningitidis Serogroup B Strains at 1 Month After the 2-dose(0,6-M) Schedule of rMenB+OMV and 1 Dose of MenACWY
Description: The effectiveness of the 2 dose (0,2-M) schedule of rMenB+OMV NZ vaccine when compared to 1 month after the MenACWY vaccination (Day 31), against a panel of N. meningitidis serogroup B strains is measured in terms of percentage of samples without bactericidal activity using enc-hSBA, which provides a qualitative assessment (yes/no) of the presence of sufficient bactericidal antibodies in human sera to kill a meningococcal strain at a specific dilution of 1:4.
Time Frame: At 1 month after the vaccination schedule (i.e., Day 91 for the MenB_0_2_6 group [2 dose schedule] and Day 31 for the MenACWY group)
Population: Analysis was performed on blood samples collected from FAS , which included all participants who were randomized, received at least 1 dose of the study treatment and had post-vaccination effectiveness data available for the specified analysis at the specified time points.
  Participants were randomly selected for testing against each strain therefore only a subset of participants were tested for each of the strains.
  Number of Participants analyzed = Total number of participants included in FAS.
Measure: Number; unit: Percentage of blood samples
Units Other Than Participants: Samples
Arm/Group | MenB_0_2_6 Group | ACWY Group
Number analyzed (Participants) | 893 | 173
Number analyzed (Samples) | 293 | 58
Percentage of blood samples
  Meningitis B M10713 Ab: number analyzed (Samples) | 266 | 45
  Meningitis B M10713 Ab | 1.9 | 15.6
  Meningitis B M08641 Ab: number analyzed (Samples) | 250 | 29
  Meningitis B M08641 Ab | 11.2 | 96.6
  Meningitis B M12898 Ab: number analyzed (Samples) | 260 | 41
  Meningitis B M12898 Ab | 12.4 | 69
  Meningitis B M09150 Ab: number analyzed (Samples) | 250 | 36
  Meningitis B M09150 Ab | 9.3 | 68.6
  Meningitis B M09401 Ab: number analyzed (Samples) | 253 | 49
  Meningitis B M09401 Ab | 47 | 98
  Meningitis B M07463 Ab: number analyzed (Samples) | 265 | 49
  Meningitis B M07463 Ab | 2.6 | 49
  Meningitis B M10496 Ab: number analyzed (Samples) | 277 | 47
  Meningitis B M10496 Ab | 50.5 | 100
  Meningitis B M14530 Ab: number analyzed (Samples) | 254 | 37
  Meningitis B M14530 Ab | 3.9 | 100
  Meningitis B M15668 Ab: number analyzed (Samples) | 252 | 49
  Meningitis B M15668 Ab | 0.4 | 87.8
  Meningitis B M14028 Ab: number analyzed (Samples) | 257 | 37
  Meningitis B M14028 Ab | 5.4 | 100
  Meningitis B M09909 Ab: number analyzed (Samples) | 266 | 42
  Meningitis B M09909 Ab | 82 | 100
  Meningitis B M14385 Ab: number analyzed (Samples) | 227 | 43
  Meningitis B M14385 Ab | 0 | 16.3
  Meningitis B M07992 Ab: number analyzed (Samples) | 249 | 36
  Meningitis B M07992 Ab | 0 | 0
  Meningitis B M09155 Ab: number analyzed (Samples) | 243 | 45
  Meningitis B M09155 Ab | 2.5 | 97.8
  Meningitis B M13085 Ab: number analyzed (Samples) | 271 | 44
  Meningitis B M13085 Ab | 21 | 66.4
  Meningitis B M18303 Ab: number analyzed (Samples) | 252 | 40
  Meningitis B M18303 Ab | 9.1 | 100
  Meningitis B M18711 Ab: number analyzed (Samples) | 261 | 33
  Meningitis B M18711 Ab | 7.7 | 75.8
  Meningitis B M15009 Ab: number analyzed (Samples) | 243 | 37
  Meningitis B M15009 Ab | 22.2 | 86.5
  Meningitis B M07773 Ab: number analyzed (Samples) | 281 | 35
  Meningitis B M07773 Ab | 1.1 | 74.3
  Meningitis B M09662 Ab: number analyzed (Samples) | 284 | 48
  Meningitis B M09662 Ab | 58.1 | 95.8
  Meningitis B M18483 Ab: number analyzed (Samples) | 234 | 37
  Meningitis B M18483 Ab | 4.3 | 77.3
  Meningitis B M11906 Ab: number analyzed (Samples) | 277 | 39
  Meningitis B M11906 Ab | 38.8 | 85.3
  Meningitis B M14987 Ab: number analyzed (Samples) | 264 | 35
  Meningitis B M14987 Ab | 10.7 | 62.3
  Meningitis B M12014 Ab: number analyzed (Samples) | 267 | 46
  Meningitis B M12014 Ab | 0.7 | 63.2
  Meningitis B M18200 Ab: number analyzed (Samples) | 241 | 47
  Meningitis B M18200 Ab | 12.1 | 34.4
  Meningitis B M08912 Ab: number analyzed (Samples) | 246 | 40
  Meningitis B M08912 Ab | 0 | 0
  Meningitis B M16748 Ab: number analyzed (Samples) | 281 | 45
  Meningitis B M16748 Ab | 0 | 0
  Meningitis B M08152 Ab: number analyzed (Samples) | 224 | 35
  Meningitis B M08152 Ab | 35.6 | 67.2
  Meningitis B M09973 Ab: number analyzed (Samples) | 271 | 48
  Meningitis B M09973 Ab | 1.5 | 83.3
  Meningitis B M15352 Ab: number analyzed (Samples) | 219 | 33
  Meningitis B M15352 Ab | 11.9 | 97
  Meningitis B M15165 Ab: number analyzed (Samples) | 265 | 42
  Meningitis B M15165 Ab | 0.8 | 92.9
  Meningitis B M08127 Ab: number analyzed (Samples) | 285 | 51
  Meningitis B M08127 Ab | 0.4 | 84.3
  Meningitis B M18347 Ab: number analyzed (Samples) | 249 | 44
  Meningitis B M18347 Ab | 60.5 | 80.4
  Meningitis B M12500 Ab: number analyzed (Samples) | 236 | 43
  Meningitis B M12500 Ab | 3.4 | 95.3
  Meningitis B M07499 Ab: number analyzed (Samples) | 259 | 51
  Meningitis B M07499 Ab | 81.1 | 100
  Meningitis B M09960 Ab: number analyzed (Samples) | 251 | 33
  Meningitis B M09960 Ab | 4.4 | 3
  Meningitis B M18045 Ab: number analyzed (Samples) | 247 | 41
  Meningitis B M18045 Ab | 0 | 92.7
  Meningitis B M10548 Ab: number analyzed (Samples) | 244 | 58
  Meningitis B M10548 Ab | 11.9 | 74.1
  Meningitis B M09354 Ab: number analyzed (Samples) | 258 | 40
  Meningitis B M09354 Ab | 0.4 | 80
  Meningitis B M11051 Ab: number analyzed (Samples) | 270 | 46
  Meningitis B M11051 Ab | 68.9 | 97.8
  Meningitis B M10104 Ab: number analyzed (Samples) | 249 | 41
  Meningitis B M10104 Ab | 61.8 | 97.6
  Meningitis B M13361 Ab: number analyzed (Samples) | 269 | 34
  Meningitis B M13361 Ab | 0.4 | 85.3
  Meningitis B M11042 Ab: number analyzed (Samples) | 210 | 43
  Meningitis B M11042 Ab | 30.1 | 84.2
  Meningitis B M18467 Ab: number analyzed (Samples) | 272 | 47
  Meningitis B M18467 Ab | 0.4 | 78.7
  Meningitis B M11113 Ab: number analyzed (Samples) | 273 | 51
  Meningitis B M11113 Ab | 43.1 | 75.6
  Meningitis B M07253 Ab: number analyzed (Samples) | 274 | 40
  Meningitis B M07253 Ab | 43.3 | 85.3
  Meningitis B M07356 Ab: number analyzed (Samples) | 247 | 29
  Meningitis B M07356 Ab | 0 | 41.4
  Meningitis B M10710 Ab: number analyzed (Samples) | 269 | 40
  Meningitis B M10710 Ab | 2.2 | 92.5
  Meningitis B M17147 Ab: number analyzed (Samples) | 274 | 41
  Meningitis B M17147 Ab | 5.1 | 100
  Meningitis B M14401 Ab: number analyzed (Samples) | 251 | 43
  Meningitis B M14401 Ab | 0.8 | 83.7
  Meningitis B M14293 Ab: number analyzed (Samples) | 264 | 47
  Meningitis B M14293 Ab | 36.4 | 95.7
  Meningitis B M08540 Ab: number analyzed (Samples) | 271 | 34
  Meningitis B M08540 Ab | 0.4 | 38.2
  Meningitis B M07960 Ab: number analyzed (Samples) | 292 | 39
  Meningitis B M07960 Ab | 4.1 | 94.9
  Meningitis B M16135 Ab: number analyzed (Samples) | 263 | 41
  Meningitis B M16135 Ab | 0.8 | 95.1
  Meningitis B M14548 Ab: number analyzed (Samples) | 286 | 38
  Meningitis B M14548 Ab | 2.8 | 94.7
  Meningitis B M09181 Ab: number analyzed (Samples) | 252 | 43
  Meningitis B M09181 Ab | 0 | 72.1
  Meningitis B M14224 Ab: number analyzed (Samples) | 268 | 40
  Meningitis B M14224 Ab | 0.7 | 82.5
  Meningitis B M07452 Ab: number analyzed (Samples) | 267 | 47
  Meningitis B M07452 Ab | 13.5 | 85.1
  Meningitis B M13520 Ab: number analyzed (Samples) | 234 | 30
  Meningitis B M13520 Ab | 0.9 | 66.7
  Meningitis B M09385 Ab: number analyzed (Samples) | 230 | 32
  Meningitis B M09385 Ab | 2.2 | 46.9
  Meningitis B M14881 Ab: number analyzed (Samples) | 258 | 40
  Meningitis B M14881 Ab | 14.7 | 95
  Meningitis B M13252 Ab: number analyzed (Samples) | 286 | 50
  Meningitis B M13252 Ab | 3.1 | 98
  Meningitis B M07818 Ab: number analyzed (Samples) | 249 | 43
  Meningitis B M07818 Ab | 0.4 | 90.7
  Meningitis B M09914 Ab: number analyzed (Samples) | 293 | 49
  Meningitis B M09914 Ab | 87.7 | 98
  Meningitis B M15083 Ab: number analyzed (Samples) | 260 | 40
  Meningitis B M15083 Ab | 63.7 | 78
  Meningitis B M11290 Ab: number analyzed (Samples) | 278 | 34
  Meningitis B M11290 Ab | 70.5 | 100
  Meningitis B M14988 Ab: number analyzed (Samples) | 251 | 40
  Meningitis B M14988 Ab | 0.4 | 60
  Meningitis B M10536 Ab: number analyzed (Samples) | 241 | 36
  Meningitis B M10536 Ab | 23.2 | 91.7
  Meningitis B M08959 Ab: number analyzed (Samples) | 267 | 47
  Meningitis B M08959 Ab | 0.4 | 85.1
  Meningitis B M08785 Ab: number analyzed (Samples) | 262 | 39
  Meningitis B M08785 Ab | 0.4 | 53.8
  Meningitis B M07245 Ab: number analyzed (Samples) | 254 | 43
  Meningitis B M07245 Ab | 0 | 23.3
  Meningitis B M19315 Ab: number analyzed (Samples) | 270 | 34
  Meningitis B M19315 Ab | 6.3 | 79.4
  Meningitis B M14376 Ab: number analyzed (Samples) | 269 | 41
  Meningitis B M14376 Ab | 0 | 92.7
  Meningitis B M08994 Ab: number analyzed (Samples) | 233 | 31
  Meningitis B M08994 Ab | 8.9 | 55.7
  Meningitis B M11646 Ab: number analyzed (Samples) | 252 | 36
  Meningitis B M11646 Ab | 1.6 | 83.3
  Meningitis B M13362 Ab: number analyzed (Samples) | 272 | 49
  Meningitis B M13362 Ab | 1.5 | 81.6
  Meningitis B M08080 Ab: number analyzed (Samples) | 244 | 45
  Meningitis B M08080 Ab | 46.8 | 87.1
  Meningitis B M08370 Ab: number analyzed (Samples) | 280 | 43
  Meningitis B M08370 Ab | 3.9 | 97.7
  Meningitis B M08129 Ab: number analyzed (Samples) | 242 | 28
  Meningitis B M08129 Ab | 7.4 | 71.4
  Meningitis B M07111 Ab: number analyzed (Samples) | 244 | 33
  Meningitis B M07111 Ab | 0.4 | 90.9
  Meningitis B M07537 Ab: number analyzed (Samples) | 253 | 47
  Meningitis B M07537 Ab | 96.4 | 100
  Meningitis B M13438 Ab: number analyzed (Samples) | 263 | 50
  Meningitis B M13438 Ab | 0.4 | 16
  Meningitis B M10661 Ab: number analyzed (Samples) | 259 | 33
  Meningitis B M10661 Ab | 2.7 | 97
  Meningitis B M10920 Ab: number analyzed (Samples) | 259 | 34
  Meningitis B M10920 Ab | 50.2 | 91.2
  Meningitis B M15564 Ab: number analyzed (Samples) | 258 | 40
  Meningitis B M15564 Ab | 0.8 | 77.5
  Meningitis B M10934 Ab: number analyzed (Samples) | 286 | 36
  Meningitis B M10934 Ab | 0 | 100
  Meningitis B M09400 Ab: number analyzed (Samples) | 261 | 39
  Meningitis B M09400 Ab | 1.1 | 97.4
  Meningitis B M08781 Ab: number analyzed (Samples) | 223 | 28
  Meningitis B M08781 Ab | 75.8 | 100
  Meningitis B M09173 Ab: number analyzed (Samples) | 244 | 42
  Meningitis B M09173 Ab | 0 | 95.2
  Meningitis B M14113 Ab: number analyzed (Samples) | 244 | 42
  Meningitis B M14113 Ab | 28.3 | 100
  Meningitis B M08389 Ab: number analyzed (Samples) | 258 | 45
  Meningitis B M08389 Ab | 1.9 | 86.7
  Meningitis B M16822 Ab: number analyzed (Samples) | 240 | 34
  Meningitis B M16822 Ab | 85 | 100
  Meningitis B M10995 Ab: number analyzed (Samples) | 282 | 47
  Meningitis B M10995 Ab | 16.3 | 85.1
  Meningitis B M08780 Ab: number analyzed (Samples) | 241 | 40
  Meningitis B M08780 Ab | 0.8 | 92.5
  Meningitis B M09910 Ab: number analyzed (Samples) | 256 | 43
  Meningitis B M09910 Ab | 1.2 | 93
  Meningitis B M08320 Ab: number analyzed (Samples) | 277 | 45
  Meningitis B M08320 Ab | 45.1 | 86.8
  Meningitis B M14879 Ab: number analyzed (Samples) | 252 | 47
  Meningitis B M14879 Ab | 3.3 | 23.2
  Meningitis B M09345 Ab: number analyzed (Samples) | 263 | 48
  Meningitis B M09345 Ab | 32.3 | 74.9
  Meningitis B M14594 Ab: number analyzed (Samples) | 254 | 44
  Meningitis B M14594 Ab | 35.8 | 97.7
  Meningitis B M07621 Ab: number analyzed (Samples) | 259 | 40
  Meningitis B M07621 Ab | 0.4 | 77.5
  Meningitis B M13568 Ab: number analyzed (Samples) | 268 | 40
  Meningitis B M13568 Ab | 9.7 | 95
  Meningitis B M18017 Ab: number analyzed (Samples) | 262 | 31
  Meningitis B M18017 Ab | 0 | 96.8
  Meningitis B M08420 Ab: number analyzed (Samples) | 260 | 40
  Meningitis B M08420 Ab | 0.8 | 95
  Meningitis B M07959 Ab: number analyzed (Samples) | 243 | 35
  Meningitis B M07959 Ab | 1.2 | 97.1
  Meningitis B M06970 Ab: number analyzed (Samples) | 243 | 32
  Meningitis B M06970 Ab | 28.8 | 90.6
  Meningitis B M10491 Ab: number analyzed (Samples) | 254 | 39
  Meningitis B M10491 Ab | 16.1 | 82.1
  Meningitis B M13569 Ab: number analyzed (Samples) | 233 | 31
  Meningitis B M13569 Ab | 0.4 | 96.8
  Meningitis B M10182 Ab: number analyzed (Samples) | 251 | 44
  Meningitis B M10182 Ab | 0 | 0
  Meningitis B M13547 Ab: number analyzed (Samples) | 260 | 44
  Meningitis B M13547 Ab | 5 | 47.7
  Meningitis B M15276 Ab: number analyzed (Samples) | 238 | 41
  Meningitis B M15276 Ab | 0.4 | 87.8

23. Secondary Outcome: Percentage of Participants Classified by Percentage of Serogroup B Invasive Disease Strains Killed Using Enc-hSBA in Each Subject at 1 Month After Vaccination Schedule for the MenB_0_2_6 Group [3 Dose], MenB_0_6 Group and Last MenABCWY Dose (Pooled Lots)
Description: The percentage of participants classified by percentage of N.meningitidis serogroup B invasive strains killed using enc-hSBA and the corresponding 2- sided 95% CI based on Clopper-Pearson method is calculated for each vaccine group. As pre-specified in the protocol, data reported in this outcome measure were presented for the MenB_0_2_6 group, MenB_0_6 group and ABCWY pooled group, participants from the ABCWY-1, ABCWY-2, and ABCWY-3 groups were pooled into a single group.
Time Frame: At 1 month after the vaccination schedule (Day 211 for MenB_0_2_6 group (3 dose schedule), MenB_0_6 group and ABCWY_Pooled group)
Population: Analysis was performed on the FAS, which included participants who were randomized, received at least 1 dose of the study treatment and had post-vaccination effectiveness data available for the specified analysis at the specified time points.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MenB_0_2_6 Group | MenB_0_6 Group | ABCWY_Pooled
Number analyzed (Participants) | 790 | 813 | 817
Percentage of participants
  >=50% killed strains | 98.7 (97.7) [97.7 to 99.4] | 98.5 (97.4) [97.4 to 99.2] | 98 (96.8) [96.8 to 98.9]
  >=55% killed strains | 98.4 (97.2) [97.2 to 99.1] | 97.4 (96.1) [96.1 to 98.4] | 96.8 (95.4) [95.4 to 97.9]
  >=60% killed strains | 97.8 (96.6) [96.6 to 98.7] | 96.8 (95.3) [95.3 to 97.9] | 95.2 (93.5) [93.5 to 96.6]
  >=65% killed strains | 96.5 (94.9) [94.9 to 97.6] | 93.6 (91.7) [91.7 to 95.2] | 90.1 (87.8) [87.8 to 92]
  >=70% killed strains | 93.4 (91.5) [91.5 to 95] | 89.8 (87.5) [87.5 to 91.8] | 84.1 (81.4) [81.4 to 86.5]
  >=75% killed strains | 86.8 (84.3) [84.3 to 89.1] | 82.2 (79.4) [79.4 to 84.7] | 74.7 (71.5) [71.5 to 77.6]
  >=80% killed strains | 79.2 (76.2) [76.2 to 82] | 75.5 (72.4) [72.4 to 78.4] | 66 (62.6) [62.6 to 69.2]
  >=85% killed strains | 62.8 (59.3) [59.3 to 66.2] | 60.4 (56.9) [56.9 to 63.8] | 50.1 (46.6) [46.6 to 53.5]
  >=90% killed strains | 43.7 (40.2) [40.2 to 47.2] | 41.3 (37.9) [37.9 to 44.8] | 32.1 (28.9) [28.9 to 35.4]
  >=95% killed strains | 22.5 (19.7) [19.7 to 25.6] | 21 (18.3) [18.3 to 24] | 13.7 (11.4) [11.4 to 16.3]
  100% killed strains | 10 (8) [8 to 12.3] | 8.4 (6.6) [6.6 to 10.5] | 6.1 (4.6) [4.6 to 8]

24. Secondary Outcome: Percentage of Participants Classified by Percentage of Serogroup B Invasive Disease Strains Killed Using Enc-hSBA in Each Subject at 1 Month After Vaccination With rMenB+OMV NZ (0,2-months)
Description: The percentage of participants classified by percentage of N.meningitidis serogroup B invasive strains killed using enc-hSBA and the corresponding 2- sided 95% CI based on Clopper-Pearson method is calculated for each vaccine group.
Time Frame: At 1 month after the vaccination schedule (Day 91 for MenB_0_2_6 group [2 dose schedule])
Population: Analysis was performed on the FAS, which included participants who were randomized, received at least 1 dose of the study treatment, and had post-vaccination effectiveness data available for the specified analysis at the specified time points.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MenB_0_2_6 Group
Number analyzed (Participants) | 831
Percentage of participants
  >=50% killed strains | 98.6 (97.5) [97.5 to 99.3]
  >=55% killed strains | 97.7 (96.5) [96.5 to 98.6]
  >=60% killed strains | 96.5 (95) [95 to 97.7]
  >=65% killed strains | 92.2 (90.1) [90.1 to 93.9]
  >=70% killed strains | 84.8 (82.2) [82.2 to 87.2]
  >=75% killed strains | 75.7 (72.6) [72.6 to 78.6]
  >=80% killed strains | 66.7 (63.3) [63.3 to 69.9]
  >=85% killed strains | 49.7 (46.2) [46.2 to 53.2]
  >=90% killed strains | 33.8 (30.6) [30.6 to 37.1]
  >=95% killed strains | 16.2 (13.8) [13.8 to 18.9]
  100% killed strains | 7.7 (6) [6 to 9.7]

25. Secondary Outcome: Percentage of Participants With hSBA Titers >= LLOQ for Each and All Serogroup B Indicator Strains at Day 1 and at 1 Month After Vaccination With rMenB+OMV NZ (0,2,6-months and 0,6-months) and Last Dose of MenABCWY (ABCWY Group-pooled Lots)
Description: The immune response to rMenB+OMV NZ and MenABCWY vaccine is evaluated by measuring bactericidal activity against each (individual response) and all (composite response) N. meningitidis serogroup B indicator strains(M14459, 96217, M13520 and NZ98/254 for fHbp, NadA, NHBA and PorA P1.4 antigens, respectively). As pre-specified in the protocol, data reported in this outcome measure were presented for the MenB_0_2_6 group, MenB_0_6 group and ABCWY pooled group, participants from the ABCWY-1, ABCWY-2, and ABCWY-3 groups were pooled into a single group.
Time Frame: At Day 1 (pre-vaccination) and1 month after the vaccination schedule (i.e., Day 211 for MenB_0_2_6 group [3 dose schedule], MenB_0_6 group and ABCWY_Pooled group)
Population: Analysis was performed on the Full Analysis Set, which included participants who were randomized, received at least 1 dose of the study treatment, and had post-vaccination effectiveness data available for the specified analysis at the specified time point.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MenB_0_2_6 Group | MenB_0_6 Group | ABCWY_Pooled
Number analyzed (Participants) | 749 | 731 | 780
Percentage of participants
  fHbp (M14459) Ab, Day 1: number analyzed (Participants) | 749 | 730 | 762
  fHbp (M14459) Ab, Day 1 | 4.9 [3.5 to 6.7] | 3.4 [2.2 to 5] | 5.4 [3.9 to 7.2]
  fHbp (M14459) Ab, Day 211: number analyzed (Participants) | 690 | 707 | 738
  fHbp (M14459) Ab, Day 211 | 97.4 [95.9 to 98.4] | 94.6 [92.7 to 96.2] | 95.9 [94.2 to 97.2]
  NadA (96217) Ab, Day 1: number analyzed (Participants) | 744 | 731 | 780
  NadA (96217) Ab, Day 1 | 6.2 [4.6 to 8.2] | 4.4 [3.0 to 6.1] | 6.2 [4.6 to 8.1]
  NadA (96217) Ab, Day 211: number analyzed (Participants) | 691 | 707 | 734
  NadA (96217) Ab, Day 211 | 100 [99.5 to 100] | 98 [96.7 to 98.9] | 96.2 [94.5 to 97.5]
  NHBA (M13520) Ab, Day 1: number analyzed (Participants) | 749 | 731 | 764
  NHBA (M13520) Ab, Day 1 | 23.2 [20.3 to 26.4] | 20.9 [18 to 24.1] | 18.5 [15.8 to 21.4]
  NHBA (M13520) Ab, Day 211: number analyzed (Participants) | 695 | 711 | 738
  NHBA (M13520) Ab, Day 211 | 97.0 [95.4 to 98.1] | 97.5 [96.0 to 98.5] | 95.3 [93.5 to 96.7]
  PorA (NZ98/254) Ab, Day 1: number analyzed (Participants) | 738 | 716 | 751
  PorA (NZ98/254) Ab, Day 1 | 2.3 [1.3 to 3.7] | 1.4 [0.7 to 2.6] | 2.1 [1.2 to 3.4]
  PorA (NZ98/254) Ab, Day 211: number analyzed (Participants) | 657 | 684 | 709
  PorA (NZ98/254) Ab, Day 211 | 85.8 [82.9 to 88.4] | 82.6 [79.5 to 85.4] | 75.3 [72.0 to 78.5]
  Composite Response, Day=1: number analyzed (Participants) | 727 | 708 | 747
  Composite Response, Day=1 | 1.1 [0.5 to 2.2] | 0.6 [0.2 to 1.4] | 1.1 [0.5 to 2.1]
  Composite Response, Day=211: number analyzed (Participants) | 654 | 683 | 707
  Composite Response, Day=211 | 83.3 [80.3 to 86.1] | 80.7 [77.5 to 83.6] | 71.4 [67.9 to 74.7]

26. Secondary Outcome: Percentage of Participants With hSBA Titers >= LLOQ for Each and All Serogroup B Indicator Strains at Day 1 and at 1 Month After Vaccination With rMenB+OMV NZ (0,2-months)
Description: The immune response to rMenB+OMV NZ is evaluated by measuring bactericidal activity against each (individual response) and all (composite response) N. meningitidis serogroup B indicator strains (M14459, 96217, M13520 and NZ98/254 for fHbp, NadA, NHBA and PorA P1.4 antigens, respectively).
Time Frame: At Day 1 (pre-vaccination) and1 month after the vaccination schedule (i.e., Day 91 for MenB_0_2_6 group [2 dose schedule])
Population: Analysis was performed on the Full Analysis Set, which included participants who were randomized, received at least 1 dose of the study treatment, and had post-vaccination effectiveness data available for the specified analysis at the specified time points.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MenB_0_2_6 Group
Number analyzed (Participants) | 753
Percentage of participants
  fHbp (M14459) Ab, Day 1: number analyzed (Participants) | 749
  fHbp (M14459) Ab, Day 1 | 4.9 [3.5 to 6.7]
  fHbp (M14459) Ab, Day 91: number analyzed (Participants) | 750
  fHbp (M14459) Ab, Day 91 | 92.9 [90.9 to 94.7]
  NadA (96217) Ab, Day 1: number analyzed (Participants) | 744
  NadA (96217) Ab, Day 1 | 6.2 [4.6 to 8.2]
  NadA (96217) Ab, Day 91 | 99.5 [98.6 to 99.9]
  NHBA, Day 1: number analyzed (Participants) | 749
  NHBA, Day 1 | 23.2 [20.3 to 26.4]
  NHBA (M13520) Ab, Day 91: number analyzed (Participants) | 750
  NHBA (M13520) Ab, Day 91 | 96.1 [94.5 to 97.4]
  PorA N (NZ98/254) Ab, Day 1: number analyzed (Participants) | 738
  PorA N (NZ98/254) Ab, Day 1 | 2.3 [1.3 to 3.7]
  PorA N (NZ98/254) Ab, Day 91: number analyzed (Participants) | 745
  PorA N (NZ98/254) Ab, Day 91 | 80 [76.9 to 82.8]
  Composite Response, Day=1: number analyzed (Participants) | 727
  Composite Response, Day=1 | 1.1 [0.5 to 2.2]
  Composite Response, Day=91: number analyzed (Participants) | 744
  Composite Response, Day=91 | 75.5 [72.3 to 78.6]

27. Secondary Outcome: Percentage of Participants With 4-fold Rise in hSBA Titers for Each of the Serogroup B Strains at 1 Month After Vaccination With rMenB+OMV NZ (0,2,6-months and 0,6-months) and Last Dose of MenABCWY (ABCWY Group-pooled Lots)
Description: The immune response to 3 dose (0,2,6-M), 2 dose (0,6-M) schedule of rMenB+OMV NZ and 2 doses of MenABCWY vaccine was evaluated by measuring bactericidal activity against each of the N. meningitidis serogroup B test strains- M14459, 96217, NZ98/254 and M13520 for fHbp, NadA, NHBA and PorA P1.4 antigens, respectively compared to baseline. Four-fold rise per each indicator strain was defined as a post-vaccination hSBA titre ≥16 for subjects with a pre-vaccination hSBA titre <4 a post-vaccination hSBA titer ≥4 times the LLOQ for subjects with a pre-vaccination hSBA titre ≥LOD and <LLOQ a post-vaccination hSBA titre ≥4 times the pre-vaccination hSBA titre for participants with a pre-vaccination hSBA titre ≥ LLOQ. As pre-specified in the protocol, data reported in this outcome measure were presented for the MenB_0_2_6 group, MenB_0_6 group and ABCWY pooled group, participants from the ABCWY-1, ABCWY-2, and ABCWY-3 groups were pooled into a single group.
Time Frame: At 1 month after the vaccination schedule (i.e., Day 211 for MenB_0_2_6 group [3 dose schedule], MenB_0_6 group and ABCWY_Pooled group) compared to Day 1 (baseline)
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MenB_0_2_6 Group | MenB_0_6 Group | ABCWY_Pooled
Number analyzed (Participants) | 685 | 704 | 731
Percentage of participants
  fHbp (M14459) Ab: number analyzed (Participants) | 679 | 699 | 729
  fHbp (M14459) Ab | 86.7 [84.0 to 89.2] | 82.4 [79.4 to 85.2] | 78.9 [75.7 to 81.8]
  NadA (96217) Ab: number analyzed (Participants) | 679 | 700 | 725
  NadA (96217) Ab | 98.7 [97.5 to 99.4] | 95.3 [93.4 to 96.7] | 92.3 [90.1 to 94.1]
  NHBA (M13520) Ab | 66.9 [63.2 to 70.4] | 69.5 [65.9 to 72.8] | 61.1 [57.5 to 64.7]
  PorA (NZ98/254) Ab: number analyzed (Participants) | 637 | 664 | 693
  PorA (NZ98/254) Ab | 56.5 [52.6 to 60.4] | 57.2 [53.4 to 61.0] | 42.4 [38.7 to 46.2]

28. Secondary Outcome: Percentage of Participants With 4-fold Rise in hSBA Titers for Each of the Serogroup B Strains at 1 Month After Vaccination With rMenB+OMV NZ (0,2 Months)
Description: The immune response to 2 dose (0,2-M) is evaluated by measuring bactericidal activity against each of the N. meningitidis serogroup B test strains- M14459, 96217, NZ98/254 and M13520 for fHbp, NadA, NHBA and PorA P1.4 antigens, respectively compared to baseline. Four-fold rise per each indicator strain was defined as a post-vaccination hSBA titre ≥16 for participants with a pre-vaccination hSBA titre <4 a post-vaccination hSBA titre ≥4 times the LLOQ for subjects with a pre-vaccination hSBA titre ≥LOD and <LLOQ a post-vaccination hSBA titre ≥4 times the pre-vaccination hSBA titre for subjects with a pre-vaccination hSBA titre ≥ LLOQ.
Time Frame: At 1 month after the vaccination schedule (i.e., Day 91 for MenB_0_2_6 [2-dose schedule]) compared to Day 1 (baseline)
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MenB_0_2_6 Group
Number analyzed (Participants) | 739
Percentage of participants
  fHbp (M14459) Ab | 74.6 [71.3 to 77.7]
  NadA (96217) Ab: number analyzed (Participants) | 738
  NadA (96217) Ab | 96.3 [94.7 to 97.6]
  NHBA (M13520) Ab | 58.5 [54.8 to 62.0]
  PorA (NZ98/254) Ab: number analyzed (Participants) | 724
  PorA (NZ98/254) Ab | 53.5 [49.7 to 57.1]

29. Secondary Outcome: hSBA Geometric Mean Titres (GMTs) Against Each of the N. Meningitidis Serogroup B Strains at Day 1 and at 1 Month After Vaccination With rMenB+OMV NZ (0,2,6-months, 0,6-months) and Last Dose of MenABCWY (ABCWY Group-pooled Lots)
Description: The immune response to rMenB+OMV NZ and MenABCWY vaccine was evaluated by measuring bactericidal activity against N. meningitidis serogroup B test strains in terms of GMTs after vaccination compared to baseline (Day 1). For each N. meningitidis serogroup B test strain (M14459, M13520, 96217 and NZ98/254 for fHbp, NadA, NHBA and PorA P1.4 antigens, respectively), The GMTs (After vaccination/baseline) are calculated, with their associated 2-sided 95% CIs. As pre-specified in the protocol, data reported in this outcome measure were presented for the MenB_0_2_6 group, MenB_0_6 group and ABCWY pooled group, participants from the ABCWY-1, ABCWY-2, and ABCWY-3 groups were pooled into a single group.
Time Frame: At Day 1 (pre-vaccination) and at 1 month after the vaccination schedule (i.e., Day 211 for MenB_0_2_6 group (3 dose schedule), MenB_0_6 group and ABCWY_Pooled group)
Population: as for outcome 26
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenB_0_2_6 Group | MenB_0_6 Group | ABCWY_Pooled
Number analyzed (Participants) | 749 | 731 | 780
Titers
  fHbp (M14459) Ab, Day 1: number analyzed (Participants) | 749 | 730 | 762
  fHbp (M14459) Ab, Day 1 | 2.8 [2.7 to 2.8] | 2.7 [2.6 to 2.8] | 2.8 [2.7 to 2.9]
  fHbp (M14459) Ab, Day 211: number analyzed (Participants) | 690 | 707 | 738
  fHbp (M14459) Ab, Day 211 | 30.8 [28.3 to 33.5] | 28.1 [25.9 to 30.6] | 25 [23 to 27.1]
  NadA (96217) Ab, Day 1: number analyzed (Participants) | 744 | 731 | 780
  NadA (96217) Ab, Day 1 | 8.4 [8.1 to 8.6] | 8.3 [8 to 8.6] | 8.5 [8.2 to 8.8]
  NadA (96217) Ab, Day 211: number analyzed (Participants) | 691 | 707 | 734
  NadA (96217) Ab, Day 211 | 267.2 [243.7 to 293] | 215.1 [196.2 to 235.9] | 150.6 [137.3 to 165.2]
  NHBA (M13520) Ab, Day 1: number analyzed (Participants) | 749 | 731 | 764
  NHBA (M13520) Ab, Day 1 | 3.4 [3.1 to 3.7] | 3.2 [3 to 3.5] | 3.1 [2.8 to 3.4]
  NHBA (M13520) Ab, Day 211: number analyzed (Participants) | 695 | 711 | 738
  NHBA (M13520) Ab, Day 211 | 30.6 [27.7 to 33.7] | 33.2 [30.2 to 36.6] | 25.2 [22.9 to 27.8]
  PorA (NZ98/254) Ab, Day 1: number analyzed (Participants) | 738 | 716 | 751
  PorA (NZ98/254) Ab, Day 1 | 3.2 [3.1 to 3.2] | 3.1 [3 to 3.2] | 3.1 [3.1 to 3.2]
  PorA (NZ98/254) Ab, Day 211: number analyzed (Participants) | 657 | 684 | 709
  PorA (NZ98/254) Ab, Day 211 | 18.1 [16.3 to 20.1] | 17.7 [15.9 to 19.6] | 12.9 [11.6 to 14.4]

30. Secondary Outcome: hSBA GMTs Against Each of the N. Meningitidis Serogroup B Strains at Day 1 and at 1 Month After Vaccination With rMenB+OMV NZ (0,2-months)
Description: The immune response to rMenB+OMV NZ and MenABCWY vaccine was evaluated by measuring bactericidal activity against N. meningitidis serogroup B test strains in terms of GMTs after vaccination compared to baseline (Day 1). For each N. meningitidis serogroup B test strain (M14459, M13520, 96217 and NZ98/254 for fHbp, NadA, NHBA and PorA P1.4 antigens, respectively), The GMTs (After vaccination/baseline) were calculated, with their associated 2-sided 95% CIs.
Time Frame: At Day 1 (pre-vaccination) and at 1 month after the vaccination schedule (i.e., Day 91 for MenB_0_2_6 group[2-dose schedule])
Population: Analysis was performed on the Full Analysis Set, which included all participants who were randomized, received at least 1 dose of the study treatment, and had post-vaccination effectiveness data available for the specified analysis at the specified time points.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenB_0_2_6 Group
Number analyzed (Participants) | 753
Titers
  fHbp (M14459) Ab, Day 1: number analyzed (Participants) | 749
  fHbp (M14459) Ab, Day 1 | 2.8 [2.7 to 2.8]
  fHbp (M14459) Ab, Day 91: number analyzed (Participants) | 750
  fHbp (M14459) Ab, Day 91 | 20.9 [18.9 to 23.1]
  NadA (96217) Ab, Day 1: number analyzed (Participants) | 744
  NadA (96217) Ab, Day 1 | 8.4 [8.1 to 8.6]
  NadA (96217) Ab, Day 91 | 178.5 [161.7 to 197.2]
  NHBA (M13520) Ab, Day 1: number analyzed (Participants) | 749
  NHBA (M13520) Ab, Day 1 | 3.4 [3.1 to 3.7]
  NHBA (M13520) Ab, Day 91: number analyzed (Participants) | 750
  NHBA (M13520) Ab, Day 91 | 27.2 [24.1 to 30.6]
  PorA (NZ98/254) Ab, Day 1: number analyzed (Participants) | 738
  PorA (NZ98/254) Ab, Day 1 | 3.2 [3.1 to 3.2]
  PorA (NZ98/254) Ab, Day 91: number analyzed (Participants) | 745
  PorA (NZ98/254) Ab, Day 91 | 17.1 [15.2 to 19.3]

31. Secondary Outcome: hSBA Geometric Mean Ratios (GMRs) for Each of the N. Meningitidis Serogroup B Strains at 1 Month After Vaccination With rMenB+OMV NZ (0,2,6-months, 0,6-months) and Last Dose of MenABCWY (ABCWY Group-pooled Lots)
Description: The immune response to rMenB+OMV NZ vaccine was evaluated by measuring bactericidal activity against N. meningitidis serogroup B test strains after vaccination compared to baseline (Day 1). For each N. meningitidis serogroup B test strain (M14459, M13520, 96217 and NZ98/254 for fHbp, NadA, NHBA and PorA P1.4 antigens, respectively), the GMRs (after vaccination/baseline) are calculated, with their associated 2-sided 95% CIs. As pre-specified in the protocol, data reported in this outcome measure were presented for the MenB_0_2_6 group, MenB_0_6 group and ABCWY pooled group, participants from the ABCWY-1, ABCWY-2, and ABCWY-3 groups were pooled into a single group.
Time Frame: At 1 month after the vaccination schedule (i.e., Day 211 for MenB_0_2_6 group (3 dose schedule), MenB_0_6 group and ABCWY_Pooled group) compared to Day 1 (baseline)
Population: as for outcome 26
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | MenB_0_2_6 Group | MenB_0_6 Group | ABCWY_Pooled
Number analyzed (Participants) | 685 | 704 | 731
Ratio
  fHbp (M14459) Ab: number analyzed (Participants) | 679 | 699 | 729
  fHbp (M14459) Ab | 11.2 [10.3 to 12.2] | 10.5 [9.6 to 11.4] | 9 [8.2 to 9.8]
  NadA (96217) Ab: number analyzed (Participants) | 679 | 700 | 725
  NadA (96217) Ab | 32.1 [29.1 to 35.3] | 25.8 [23.5 to 28.4] | 17.7 [16 to 19.4]
  NHBA (M13520) Ab | 9.1 [8.2 to 10.1] | 10.6 [9.5 to 11.7] | 8.2 [7.4 to 9.1]
  PorA (NZ98/254) Ab: number analyzed (Participants) | 637 | 664 | 693
  PorA (NZ98/254) Ab | 5.8 [5.2 to 6.5] | 5.8 [5.2 to 6.4] | 4.1 [3.7 to 4.6]

32. Secondary Outcome: hSBA GMRs for Each of the N. Meningitidis Serogroup B Strains at 1 Month After Vaccination With rMenB+OMV NZ (0,2-months)
Description: The immune response to rMenB+OMV NZ vaccine was evaluated by measuring bactericidal activity against N. meningitidis serogroup B test strains after vaccination compared to baseline (Day 1). For each N. meningitidis serogroup B test strain (M14459, M13520, 96217 and NZ98/254 for fHbp, NadA, NHBA and PorA P1.4 antigens, respectively), the GMRs (after vaccination/baseline) are calculated, with their associated 2-sided 95% CIs.
Time Frame: At 1 month after the vaccination schedule (i.e., Day 91 for MenB_0_2_6 group [2-dose schedule]) compared to Day 1 (baseline)
Population: as for outcome 26
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | MenB_0_2_6 Group
Number analyzed (Participants) | 739
Ratio
  fHbp (M14459) Ab | 7.7 [6.9 to 8.5]
  NadA (96217) Ab: number analyzed (Participants) | 738
  NadA (96217) Ab | 21.7 [19.5 to 24]
  NHBA (M13520) Ab | 8 [7.1 to 9]
  PorA (NZ98/254) Ab: number analyzed (Participants) | 724
  PorA (NZ98/254) Ab | 5.5 [4.9 to 6.2]

33. Secondary Outcome: Percentage of Participants With hSBA Titers >= LLOQ for Each of the N. Meningitidis Serogroups A,C,W,Y at Day 1 and at 1 Month After the First and the Last MenABCWY Vaccination for ABCWY_Pooled Group and 1 Month After the MenACWY Vaccine for ACWY Group
Description: The immune responses to MenABCWY and MenACWY vaccines were evaluated by measuring bactericidal activity against N. meningitidis serogroups A, C, W and Y after vaccination compared to baseline (Day 1) and expressed as the percentage of participants with hSBA titers >= LLOQ for serogroups A, C, W and Y at baseline and 1 month after vaccination schedule of MenABCWY and MenACWY vaccines. As pre-specified in the protocol, data reported in this outcome measure were presented for the ACWY group and ABCWY pooled group, participants from the ABCWY-1, ABCWY-2, and ABCWY-3 groups were pooled into a single group.
Time Frame: At Day 1, and 1 month after vaccination schedule (i.e, at Day 31 for ABCWY group [pooled lots -first dose] and for ACWY Group, and at Day 211 for ABCWY group [pooled lots - second dose])
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ABCWY_Pooled | ACWY Group
Number analyzed (Participants) | 1489 | 141
Percentage of participants
  Men A, Day 1: number analyzed (Participants) | 1452 | 137
  Men A, Day 1 | 9.2 [7.7 to 10.8] | 11.7 [6.8 to 18.3]
  Men A, Day 31: number analyzed (Participants) | 132 | 133
  Men A, Day 31 | 79.5 [71.7 to 86.1] | 90.2 [83.9 to 94.7]
  Men A, Day 211: number analyzed (Participants) | 1446 | 0
  Men A, Day 211 | 98.6 [97.9 to 99.2] |
  Men C, Day 1: number analyzed (Participants) | 1487 | 139
  Men C, Day 1 | 29.8 [27.5 to 32.2] | 28.8 [21.4 to 37.1]
  Men C, Day 31: number analyzed (Participants) | 139 | 136
  Men C, Day 31 | 74.8 [66.8 to 81.8] | 64.0 [55.3 to 72.0]
  Men C, Day 211: number analyzed (Participants) | 1457 | 0
  Men C, Day 211 | 99.6 [99.1 to 99.8] |
  Men W, Day 1: number analyzed (Participants) | 1473 | 140
  Men W, Day 1 | 12.6 [10.9 to 14.4] | 12.9 [7.8 to 19.6]
  Men W, Day 31: number analyzed (Participants) | 142 | 137
  Men W, Day 31 | 80.3 [72.8 to 86.5] | 69.3 [60.9 to 76.9]
  Men W, Day 211: number analyzed (Participants) | 1463 | 0
  Men W, Day 211 | 99.2 [98.7 to 99.6] |
  Men Y, Day 1 | 12.2 [10.6 to 14.0] | 13.5 [8.3 to 20.2]
  Men Y, Day 31: number analyzed (Participants) | 146 | 140
  Men Y, Day 31 | 82.2 [75.0 to 88.0] | 80.0 [72.4 to 86.3]
  Men Y, Day 211: number analyzed (Participants) | 1461 | 0
  Men Y, Day 211 | 99.2 [98.7 to 99.6] |

34. Secondary Outcome: Percentage of Participants With 4-fold Rise in hSBA Titers for Each of the N. Meningitidis Serogroups A, C, W and Y at 1 Month After the First MenABCWY Dose for ABCWY_Pooled Group Compared to the MenACWY Vaccine for ACWY Group Relative to Baseline (Day 1)
Description: The immune response to MenABCWY vaccine compared to MenACWY vaccine was evaluated by measuring bactericidal activity against each of the N. meningitidis serogroups A, C, W and Y at Day 31 compared to baseline (Day 1).
  Four-fold rise is defined as:
  - If the pre-vaccination hSBA titer is < 4, then post-vaccination hSBA titer should be ≥ 16. - If the pre-vaccination hSBA titer is ≥ LOD but < LLOQ, then post-vaccination hSBA titer should be ≥ 4 times the LLOQ. - If the pre-vaccination hSBA titer is ≥ LLOQ, then post-vaccination hSBA titer should be ≥ 4 times the pre-vaccination hSBA titer. The corresponding 2- sided 95% CI based on Clopper-Pearson method is calculated for each vaccine group. As pre-specified in the protocol, data reported in this outcome measure were presented for the ACWY group and ABCWY pooled group, participants from the ABCWY-1, ABCWY-2, and ABCWY-3 groups were pooled into a single group.
Time Frame: At 1 month after vaccination schedule (i.e, at Day 31 for ABCWY group [pooled group] and for ACWY Group) relative to baseline (Day 1)
Population: Analysis was performed on the Full Analysis Set, which included participants who were randomized, received at least 1 dose of the study treatment, and had post-vaccination effectiveness available for the specified analysis at the specified time points.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ABCWY_Pooled | ACWY Group
Number analyzed (Participants) | 146 | 140
Percentage of participants
  Men A: number analyzed (Participants) | 127 | 129
  Men A | 74.0 [65.5 to 81.4] | 86.0 [78.8 to 91.5]
  Men C: number analyzed (Participants) | 139 | 134
  Men C | 66.9 [58.4 to 74.6] | 56.7 [47.9 to 65.2]
  Men W: number analyzed (Participants) | 139 | 136
  Men W | 74.1 [66.0 to 81.2] | 66.2 [57.6 to 74.1]
  Men Y | 76.0 [68.3 to 82.7] | 72.1 [63.9 to 79.4]

35. Secondary Outcome: hSBA GMTs Against Each of the N. Meningitidis Serogroups A, C, W and Y at Day 1 and 1 Month After the First and the Last MenABCWY Vaccination for the ABCWY_Pooled Group and at 1 Month After the MenACWY Vaccination for ACWY Group
Description: The immune responses to MenABCWY and MenACWY vaccines are evaluated by measuring bactericidal activity against N. meningitidis serogroups A, C, W and Y in terms of GMTs after vaccination compared to baseline (Day 1). For each N. meningitidis serogroups A, C, W and Y, the GMTs (after vaccination/baseline) are calculated, with their associated 2-sided 95% CIs. As pre-specified in the protocol, data reported in this outcome measure were presented for the ACWY group and ABCWY pooled group, participants from the ABCWY-1, ABCWY-2, and ABCWY-3 groups were pooled into a single group.
Time Frame: as for outcome 33
Population: as for outcome 26
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | ABCWY_Pooled | ACWY Group
Number analyzed (Participants) | 1489 | 141
Titers
  Men A, Day 1: number analyzed (Participants) | 1452 | 137
  Men A, Day 1 | 11.1 [10.3 to 11.9] | 12.7 [10.9 to 14.8]
  Men A, Day 31: number analyzed (Participants) | 132 | 133
  Men A, Day 31 | 175.3 [121.2 to 253.3] | 474.8 [331.3 to 680.3]
  Men A, Day 211: number analyzed (Participants) | 1446 | 0
  Men A, Day 211 | 352.0 [322.0 to 384.7] |
  Men C, Day 1: number analyzed (Participants) | 1487 | 139
  Men C, Day 1 | 12.0 [10.9 to 13.3] | 11.4 [9.1 to 14.3]
  Men C, Day 31: number analyzed (Participants) | 139 | 136
  Men C, Day 31 | 674.8 [355.9 to 1279.4] | 379.0 [204.4 to 703.0]
  Men C, Day 211: number analyzed (Participants) | 1457 | 0
  Men C, Day 211 | 1162.5 [1015.7 to 1330.5] |
  Men W, Day 1: number analyzed (Participants) | 1473 | 140
  Men W, Day 1 | 8.0 [7.4 to 8.7] | 7.4 [6.2 to 8.9]
  Men W, Day 31: number analyzed (Participants) | 142 | 137
  Men W, Day 31 | 374.0 [243.4 to 574.8] | 194.3 [128.3 to 294.2]
  Men W, Day 211: number analyzed (Participants) | 1463 | 0
  Men W, Day 211 | 666.5 [603.2 to 736.3] |
  Men Y, Day 1 | 9.3 [8.7 to 10.0] | 9.9 [8.6 to 11.5]
  Men Y, Day 31: number analyzed (Participants) | 146 | 140
  Men Y, Day 31 | 375.4 [246.9 to 570.7] | 320.9 [213.8 to 481.7]
  Men Y, Day 211: number analyzed (Participants) | 1461 | 0
  Men Y, Day 211 | 655.9 [587.0 to 733.0] |

36. Secondary Outcome: GMRs for Each of the N. Meningitidis Serogroups A, C, W and Y at 1 Month After the First and the Last MenABCWY Vaccination for the ABCWY _Pooled Group and at 1 Month After the MenACWY Vaccination for ACWY Group
Description: The immune responses to MenABCWY and MenACWY vaccines are evaluated by measuring bactericidal activity against N. meningitidis serogroups A, C, W and Y. For each N. meningitidis serogroups A, C, W and Y, the GMRs (after vaccination/baseline) are calculated, with their associated 2-sided 95% CIs. As pre-specified in the protocol, data reported in this outcome measure were presented for the ACWY group and ABCWY pooled group, participants from the ABCWY-1, ABCWY-2, and ABCWY-3 groups were pooled into a single group.
Time Frame: 1 month after vaccination schedule (i.e, at Day 31 for ABCWY group [pooled lots -first dose] and for ACWY Group, and at Day 211 for ABCWY group [pooled lots - second dose]) compared to baseline (Day 1)
Population: as for outcome 26
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | ABCWY_Pooled | ACWY Group
Number analyzed (Participants) | 1446 | 140
Ratio
  Men A, Day 31: number analyzed (Participants) | 127 | 129
  Men A, Day 31 | 11.8 [7.9 to 17.7] | 31.8 [21.4 to 47.1]
  Men A, Day 211: number analyzed (Participants) | 1397 | 0
  Men A, Day 211 | 31.2 [28.3 to 34.5] |
  Men C, Day 31: number analyzed (Participants) | 139 | 134
  Men C, Day 31 | 30.9 [16.9 to 56.2] | 22.9 [12.8 to 41.1]
  Men C, Day 211: number analyzed (Participants) | 1439 | 0
  Men C, Day 211 | 96.9 [84.5 to 111.1] |
  Men W, Day 31: number analyzed (Participants) | 139 | 136
  Men W, Day 31 | 32.9 [21.7 to 50.0] | 23.2 [15.5 to 34.7]
  Men W, Day 211: number analyzed (Participants) | 1432 | 0
  Men W, Day 211 | 83.8 [74.9 to 93.8] |
  Men Y, Day 31: number analyzed (Participants) | 146 | 140
  Men Y, Day 31 | 28.1 [18.3 to 43.2] | 25.6 [16.9 to 38.8]
  Men Y, Day 211: number analyzed (Participants) | 1446 | 0
  Men Y, Day 211 | 70.2 [62.3 to 79.1] |

37. Secondary Outcome: Total Immunoglobulin G (IgG) Antibodies Concentrations Against N. Meningitidis Serogroups A, C, W and Y at Day 1 and 1 Month After the First and the Last MenABCWY Vaccination for ABCWY _Pooled Group and 1 Month After the MenACWY Vaccination for ACWY Group
Description: The immune responses to MenABCWY and MenACWY vaccines were evaluated by measuring the total IgG in terms of electrochemiluminescence-based multiplex (ECL) geometric mean concentrations (GMCs) which was an alternative assay to Enzyme-Linked Immunosorbent Assay (ELISA). ECL (validated assay) was used because ELISA is not validated. As pre- specified in the protocol, data reported in this outcome measure were presented for the ACWY group and ABCWY pooled group, participants from the ABCWY-1, ABCWY-2, and ABCWY-3 groups were pooled into a single group.
Time Frame: as for outcome 33
Population: as for outcome 26
Measure: Geometric Mean (95% Confidence Interval); unit: microgram per milliliter(µg/mL)
Arm/Group | ACWY Group | ABCWY_Pooled
Number analyzed (Participants) | 172 | 179
microgram per milliliter(µg/mL)
  Men A, Day 1: number analyzed (Participants) | 170 | 179
  Men A, Day 1 | 2.3 [2.0 to 2.7] | 1.9 [1.6 to 2.2]
  Men A, Day 31: number analyzed (Participants) | 168 | 177
  Men A, Day 31 | 53.7 [40.8 to 70.7] | 18.1 [13.8 to 23.8]
  Men A, Day 211: number analyzed (Participants) | 0 | 164
  Men A, Day 211 |  | 30.2 [23.3 to 39.2]
  Men C, Day 1: number analyzed (Participants) | 170 | 179
  Men C, Day 1 | 0.8 [0.7 to 1.0] | 0.7 [0.6 to 0.8]
  Men C, Day 31: number analyzed (Participants) | 170 | 175
  Men C, Day 31 | 13.8 [10.4 to 18.4] | 15.5 [11.6 to 20.7]
  Men C, Day 211: number analyzed (Participants) | 0 | 163
  Men C, Day 211 |  | 17.0 [13.1 to 22.0]
  Men W, Day 1: number analyzed (Participants) | 170 | 179
  Men W, Day 1 | 0.6 [0.5 to 0.7] | 0.5 [0.4 to 0.6]
  Men W, Day 31: number analyzed (Participants) | 172 | 178
  Men W, Day 31 | 8.4 [6.0 to 11.6] | 9.1 [6.5 to 12.8]
  Men W, Day 211: number analyzed (Participants) | 0 | 164
  Men W, Day 211 |  | 21.7 [16.0 to 29.5]
  Men Y, Day 1: number analyzed (Participants) | 170 | 179
  Men Y, Day 1 | 0.9 [0.8 to 1.0] | 0.9 [0.7 to 1.0]
  Men Y, Day 31: number analyzed (Participants) | 172 | 178
  Men Y, Day 31 | 14.3 [10.2 to 19.8] | 12.9 [9.2 to 18.0]
  Men Y, Day 211: number analyzed (Participants) | 0 | 164
  Men Y, Day 211 |  | 26.3 [19.6 to 35.4]

ADVERSE EVENTS:
Time Frame: SAEs and Non-serious AEs (Other AEs) were collected through the entire period of the study (from Day 1 up to study end [Day 361])
Arm/Group | MenB_0_2_6 Group | MenB_0_6 Group | ACWY Group | ABCWY-1 Group | ABCWY-2 Group | ABCWY-3 Group
All-Cause Mortality (participants affected / at risk) | 1/897 | 1/906 | 0/178 | 0/549 | 0/554 | 0/554
Serious Adverse Events (participants affected / at risk) | 20/897 | 22/906 | 5/178 | 8/549 | 9/554 | 8/554
Other Adverse Events (participants affected / at risk) | 876/897 | 872/906 | 173/178 | 529/549 | 537/554 | 544/554
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | MenB_0_2_6 Group (N=897) | MenB_0_6 Group (N=906) | ACWY Group (N=178) | ABCWY-1 Group (N=549) | ABCWY-2 Group (N=554) | ABCWY-3 Group (N=554)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urachal abnormality (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypermetropia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis toxic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected dermal cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post-acute COVID-19 syndrome (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic liver injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin T increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain stem glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ovarian fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0) | 0/0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuromyelitis optica spectrum disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paresis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petit mal epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Speech disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Complication of pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Placental insufficiency (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorexia nervosa (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression suicidal (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0/0 (0) | 1/1 (1) | 0/0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Substance-induced psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thinking abnormal (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vancomycin infusion reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | MenB_0_2_6 Group (N=897) | MenB_0_6 Group (N=906) | ACWY Group (N=178) | ABCWY-1 Group (N=549) | ABCWY-2 Group (N=554) | ABCWY-3 Group (N=554)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 5 (6) | 7 (7) | 1 (1) | 4 (4) | 2 (2) | 3 (3)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Tachycardia paroxysmal (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0/540 (0) | 0 (0) | 0 (0)
Dermoid cyst (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Familial mediterranean fever (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple endocrine neoplasia Type 1 (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pectus excavatum (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rathke's cleft cyst (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type V hyperlipidaemia (Congenital, familial and genetic disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Ear discomfort (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 3 (3) | 2 (2) | 0 (0) | 2 (2) | 3 (3) | 1 (1)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Excessive cerumen production (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
External ear inflammation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Motion sickness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tympanosclerosis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 4 (4) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Growth hormone deficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thyroid cyst (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thyroid stimulating hormone deficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Astigmatism (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blindness transient (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chalazion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye inflammation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye irritation (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye swelling (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid exfoliation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eyelid ptosis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Swelling of eyelid (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 11 (12) | 1 (1) | 6 (7) | 3 (3) | 4 (7)
Abdominal pain lower (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 7 (7) | 9 (10) | 2 (2) | 6 (6) | 3 (4) | 9 (10)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coeliac disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 14 (15) | 16 (19) | 5 (5) | 6 (6) | 4 (4) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 2 (2)
Embedded tooth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Gastritis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 4 (4) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperchlorhydria (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lip swelling (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 245 (324) | 204 (262) | 45 (59) | 121 (156) | 138 (174) | 139 (170)
Oral pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral pruritus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palatal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis relapsing (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue discolouration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 5 (6) | 1 (1) | 3 (3) | 2 (2) | 2 (2)
Transient lingual papillitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (6) | 11 (11) | 1 (1) | 2 (2) | 6 (6) | 4 (4)
Administration site erythema (General disorders) | 209 (300) | 157 (203) | 21 (24) | 112 (134) | 115 (143) | 94 (120)
Administration site induration (General disorders) | 138 (180) | 113 (142) | 17 (19) | 73 (93) | 78 (92) | 72 (88)
Administration site pain (General disorders) | 851 (2229) | 853 (1768) | 149 (240) | 515 (1003) | 522 (1025) | 524 (1028)
Administration site swelling (General disorders) | 202 (293) | 158 (200) | 22 (25) | 101 (134) | 109 (146) | 95 (121)
Asthenia (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Chills (General disorders) | 8 (8) | 3 (4) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Cyst (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 604 (1183) | 579 (1005) | 105 (174) | 352 (601) | 356 (609) | 358 (597)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Induration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 2 (2) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Injection site bruising (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Injection site discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site eczema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site haematoma (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site hypoaesthesia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site induration (General disorders) | 8 (11) | 5 (5) | 2 (2) | 3 (4) | 5 (5) | 5 (5)
Injection site mass (General disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Injection site pain (General disorders) | 3 (3) | 8 (8) | 1 (1) | 5 (5) | 5 (5) | 3 (3)
Injection site papule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site paraesthesia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Injection site pruritus (General disorders) | 2 (4) | 1 (2) | 1 (1) | 0 (0) | 2 (3) | 3 (3)
Injection site rash (General disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site warmth (General disorders) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Malaise (General disorders) | 4 (5) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Medical device pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 4 (5) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 66 (69) | 59 (62) | 7 (7) | 37 (41) | 46 (49) | 32 (32)
Swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Swelling face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thirst (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaccination site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaccination site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination site pruritus (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaccination site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaccination site urticaria (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination site warmth (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vessel puncture site pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Allergy to animal (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allergy to arthropod sting (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaphylactoid reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dust allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Food allergy (Immune system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multiple allergies (Immune system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 7 (7) | 7 (7) | 2 (2) | 2 (2) | 1 (1) | 6 (6)
Acarodermatitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Adenovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asymptomatic COVID-19 (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Body tinea (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Bullous impetigo (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 93 (96) | 107 (111) | 26 (26) | 63 (63) | 71 (71) | 61 (64)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chlamydial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 4 (4)
Conjunctivitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronavirus infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 4 (4) | 0 (0)
Ear infection (Infections and infestations) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Ear lobe infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Endometritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterobiasis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema migrans (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fungal foot infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 6 (6) | 4 (5) | 0 (0) | 5/540 (5) | 6 (6) | 5 (5)
Gastroenteritis viral (Infections and infestations) | 3 (3) | 6 (6) | 0 (0) | 2 (2) | 3 (3) | 2 (2)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Genital herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Helminthic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Impetigo (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Infected bite (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 10 (10) | 11 (12) | 1 (1) | 10 (10) | 5 (5) | 7 (7)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Laryngotracheitis obstructive (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lyme disease (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Molluscum contagiosum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mycoplasma genitalium infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 29 (33) | 37 (42) | 11 (11) | 16 (17) | 20 (21) | 24 (27)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 5 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 4 (5) | 4 (4) | 0 (0) | 4 (4) | 5 (5) | 1 (1)
Otitis media (Infections and infestations) | 6 (6) | 3 (3) | 0 (0) | 4 (4) | 1 (1) | 1 (1)
Otitis media acute (Infections and infestations) | 3 (4) | 1 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Otosalpingitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parasitic gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Parotitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericoronitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 8 (9) | 19 (24) | 2 (2) | 10 (12) | 9 (9) | 9 (9)
Pharyngitis streptococcal (Infections and infestations) | 2 (2) | 4 (4) | 1 (1) | 1 (1) | 4 (4) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post-acute COVID-19 syndrome (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulpitis dental (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 2 (3) | 7 (8) | 2 (2) | 3 (4) | 4 (4) | 4 (6)
Rhinitis (Infections and infestations) | 4 (4) | 8 (8) | 2 (2) | 2 (2) | 2 (2) | 2 (2)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sialoadenitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 4 (4) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Skin bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Streptococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suspected COVID-19 (Infections and infestations) | 5 (5) | 6 (6) | 0 (0) | 2 (2) | 3 (3) | 5 (6)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinea versicolour (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tonsillitis (Infections and infestations) | 10 (10) | 15 (17) | 5 (6) | 4 (5) | 2 (3) | 14 (14)
Tonsillitis streptococcal (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trichomoniasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 35 (38) | 42 (46) | 6 (6) | 24 (25) | 22 (23) | 25 (26)
Upper respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 9 (11) | 9 (10) | 3 (3) | 6 (10) | 4 (4) | 3 (3)
Vaccination site cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaccination site pustule (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Varicella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 4 (5) | 5 (6) | 0 (0) | 2 (2) | 4 (5) | 1 (1)
Viral pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 3 (3) | 4 (4) | 0 (0) | 6 (6) | 0 (0) | 3 (3)
Vulvovaginal candidiasis (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Vulvovaginitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Yersinia infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaesthetic complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Animal scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bursa injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 0 (0) | 2 (3) | 4 (4) | 2 (5)
Ear canal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 2 (2) | 5 (6) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Foreign body in respiratory tract (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 1 (2)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Human bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 4 (4) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 5 (7) | 16 (17) | 1 (1) | 5 (5) | 4 (4) | 5 (5)
Limb crushing injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 3 (3) | 5 (5) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0/0 (0) | 1/1 (1) | 0/0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle rupture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Musculoskeletal foreign body (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nail injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural dizziness (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Procedural vomiting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scratch (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 3 (3) | 2 (3) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 5 (5) | 5 (5) | 1 (1) | 0 (0) | 3 (3) | 2 (2)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sports injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stress fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tooth injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Torus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0) | 4 (4) | 3 (3) | 2 (2)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Computerised tomogram abdomen abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heart rate irregular (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Red blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 6 (6) | 7 (7) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
Serum ferritin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Streptococcus test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroid hormones decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Folate deficiency (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gluten sensitivity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haemochromatosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypovitaminosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insulin resistance (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Lactose intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin B complex deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Zinc deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 154 (205) | 127 (163) | 25 (30) | 84 (105) | 76 (95) | 76 (90)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Axillary mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 15 (15) | 2 (2) | 5 (5) | 8 (8) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Epiphysiolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Growing pains (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint hyperextension (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint warmth (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Knee deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 240 (325) | 209 (276) | 30 (35) | 122 (153) | 132 (178) | 130 (169)
Myokymia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 11 (11) | 1 (1) | 2 (2) | 2 (2) | 5 (8)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sever's disease (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Short stature (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal flattening (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Torticollis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign soft tissue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 6 (8) | 6 (6) | 1 (1) | 1 (1) | 3 (3) | 3 (3)
Dyskinesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 578 (999) | 525 (874) | 97 (148) | 300 (512) | 309 (525) | 320 (541)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 3 (3) | 5 (5) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Myoclonus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Neuromuscular blockade (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Psychomotor hyperactivity (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep deficit (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Speech disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 7 (7)
Taste disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Acute stress disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adjustment disorder (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anger (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anorexia nervosa (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 6 (6) | 8 (8) | 0 (0) | 6 (6) | 2 (2) | 3 (3)
Anxiety disorder (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Binge eating (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 6 (6) | 4 (4) | 2 (2) | 4 (4) | 6 (6) | 4 (4)
Depression suicidal (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disruptive mood dysregulation disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 5 (5)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mixed anxiety and depressive disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Obsessive-compulsive disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
School refusal (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stress (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tic (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (3)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephritis (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract inflammation (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Amenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bartholin's cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast haematoma (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast inflammation (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast tenderness (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 14 (19) | 10 (10) | 6 (6) | 9 (11) | 6 (6) | 10 (14)
Endometriosis (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Menstruation delayed (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nipple enlargement (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Penile rash (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Premenstrual pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Premenstrual syndrome (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine spasm (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 6 (8) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (4) | 3 (3) | 2 (2) | 7 (7) | 7 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 12 (13) | 6 (6) | 0 (0) | 6 (8) | 3 (3) | 7 (7)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 11 (12) | 0 (0) | 13 (13) | 7 (7) | 9 (9)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 2 (2) | 3 (3) | 4 (4) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Throat clearing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillolith (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 8 (8) | 7 (7) | 1 (1) | 6 (7) | 2 (2) | 4 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cold urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 1 (2)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2) | 0 (0) | 2 (3) | 1 (1) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pityriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 0 (0) | 7 (7) | 2 (2) | 4 (4)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin induration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Urticaria chronic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Menarche (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperaemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pallor (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral venous disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-05-12): https://cdn.clinicaltrials.gov/large-docs/93/NCT04502693/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-06): https://cdn.clinicaltrials.gov/large-docs/93/NCT04502693/SAP_002.pdf